## Statistical Analysis Plan

# Allakos, Inc Protocol AK001-002

# A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate Multiple Doses of AK001 in Patients With Moderate to Severe Nasal Polyposis

**VERSION 1.0 DATED 16 August 2017** 

Sponsor: Allakos, Inc.

75 Shoreway Road, Suite A San Carlos, CA 94070

Prepared by: Mojtaba Noursalehi, Ph.D.

InClin, Inc.

2000 Alameda De Las Pulgas

San Mateo, CA 94403

**Version:** 1, 16 August 2017

# Approval

Upon review of this document, including table, listing, and figure shells, the undersigned approves the Statistical Analysis Plan. The analysis methods and data presentation are acceptable.

| Signature | Date |
|---|---|
| Matthew P. Kovalsky Senior Director, Clinical Operations Allakos, Inc. | 16 As6 2017 |
| Mojtaba Noursalehi, PhD<br>SVP, Biometrics Consultant<br>InClin, Inc. | 17 AUB 201. |

## **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 10 |
|----|---------------------------------------------------------------|----|
| | 1.1 General | 10 |
| | 1.2 PROTOCOL VERSIONS | 10 |
| 2. | STUDY OBJECTIVES | 10 |
| 3. | STUDY DESIGN | 12 |
| 4. | DETERMINATION OF SAMPLE SIZE | 13 |
| 5. | GENERAL ANALYSIS CONSIDERATIONS | 14 |
| | 5.1 CONVENTIONS | 15 |
| | 5.2 STANDARD CALCULATIONS | |
| | 5.3 HANDLING PARTIAL DATES FOR ADVERSE EVENTS AND MEDICATIONS | |
| | 5.4 VISIT WINDOWS | |
| | 5.5 REVIEW OF BLINDED DATA | 18 |
| 6. | ANALYSIS POPULATIONS | 18 |
| 7. | STUDY POPULATION | 19 |
| | 7.1 SUBJECT DISPOSITION | |
| | 7.2 Protocol Deviations | |
| | 7.3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS | |
| | 7.4 MEDICAL HISTORY | |
| | 7.5 PHYSICAL EXAMINATIONS | 20 |
| | 7.6 VITAL SIGNS | |
| | 7.7 ECG | |
| | 7.8 FECAL COLLECTION | |
| | 7.9 Adverse Events | |
| | 7.10 Laboratory Values | |
| | 7.11 ANTI-DRUG ANTIBODY (ADA) | |
| | 7.12 PRIOR AND CONCOMITANT MEDICATIONS | |
| 8. | EFFICACY ANALYSES | |
| | 8.1 Efficacy Variables | |
| | 8.1.1 Primary Efficacy Variable | |
| | 8.1.2 SECONDARY EFFICACY VARIABLES | |
| | 8.1.3 EXPLORATORY EFFICACY VARIABLES | |
| | 8.2 ADJUSTMENTS FOR COVARIATES | |
| | 8.3 HANDLING OF DROPOUTS OR MISSING DATA | |
| | 8.4 INTERIM ANALYSIS AND DATA MONITORING | |
| | 8.5 EXAMINATION OF SUBGROUPS | |
| | 8.6 MULTIPLE COMPARISONS/MULTIPLICITY | |
| _ | 8.7 MULTICENTER STUDIES | |
| 9 | METHODS OF EFFICACY ANALYSIS | 26 |

| | 9.1 Primary Efficacy Analyses | 26 |
|---|---|---|
| | 9.2 SENSITIVITY EFFICACY ANALYSES OF PRIMARY ENDPOINTS | 27 |
| | 9.2.1 ANALYSIS FOR TPS IN PRESENCE OF MISSING DATA | 27 |
| | 9.2.2 THE ANALYSIS WITH TPS INCLUDING TIME AS A REPEATED FACTOR | 28 |
| | 9.2.3 ANALYSIS OF TPS IN ABSOLUTE VALUE AND PERCENT CHANGE FROM BASELINE | 28 |
| | 9.2.4 ALTERNATE ANALYSIS POPULATION | |
| | 9.2.5 TIME TO RESPONSE. | 28 |
| | 9.2.6 SUBGROUP ANALYSES | |
| | 9.3 SECONDARY EFFICACY ANALYSES | |
| | 9.4 EXPLORATORY EFFICACY ANALYSES | |
| | 9.5 PHARMACOKINETIC AND BIOMARKER ANALYSES | 31 |
| 10. | SAFETY ANALYSES | 32 |
| | 10.1 Adverse Events | 33 |
| | 10.1.1 SELECTED SUBSETS OF ADVERSE EVENTS | 34 |
| | 10.1.2 SUBGROUP ANALYSES. | 34 |
| | 10.2 CLINICAL LABORATORY EVALUATION | 34 |
| | 10.3 VITAL SIGNS | |
| | 10.4 PRIOR AND CONCOMITANT MEDICATIONS | 37 |
| 11. | CHANGES TO PROTOCOL-SPECIFIED ANALYSES | 37 |
| 12. | REFERENCES | 37 |
| ΑP | PENDICES | 39 |
| | APPENDIX A: VISIT WINDOWS | |
| | APPENDIX B: CRITERIA FOR DETERMINING POTENTIALLY CLINICALLY SIGNIFICANT | 57 |
| | VALUES IN LABORATORY TEST RESULTS | 40 |
| | APPENDIX C: CRITERIA FOR DETERMINING POTENTIALLY CLINICALLY SIGNIFICANT | |
| | VALUES IN VITAL SIGNS | 42 |
| | APPENDIX D: CRITERIA FOR IDENTIFYING ECG VALUES THAT REFLECT POTENTIALLY | |
| | CLINICALLY SIGNIFICANT CHANGE | 43 |
| | APPENDIX E: RULES FOR DETERMINING "WORST" VALUE | 44 |
| | APPENDIX F: RULES FOR SCORING THE DISEASE ASSESSMENT SCALES | 45 |
| | 1. TPS | |
| | 2. THE LUND-MACKAY SCORING SYSTEM | |
| | 3. University of Pennsylvania Smell Identification Test <sup>tm</sup> | |
| | 4. SINO-NASAL OUTCOME TEST-22 | 47 |
| | 5. VISUAL ANALOGUE SCALES FOR SYMPTOMS OF RHINOSINUSITIS AND CLINICAL | |
| | SYMPTOMS IMPROVEMENT SCALE | |
| | 6. 36-ITEM SHORT FORM HEALTH SURVEY | |
| | 7. ASTHMA CONTROL TEST <sup>TM</sup> | |
| | APPENDIX G: LIST OF REVIEW FILES PROVIDED BY ALLAKOS TO INCLIN | |
| | APPENDIX H: LIST OF TABLES, FIGURES, AND LISTINGS | |
| | LIST OF TABLES. | |
| | LIST OF FIGURES | 65 |

| LIST OF DATA LISTINGS | 66 |
|-----------------------------|-----|
| APPENDIX I: TABLE LAYOUTS | |
| APPENDIX J: FIGURE LAYOUTS | 131 |
| APPENDIX K. LISTING LAYOUTS | 135 |

| LIST OF ABBREVIATIONS | |
|---|---|
| ACT | Asthma Control Test <sup>TM</sup> |
| ADA | Anti-drug Antibody |
| AE | Adverse Event |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| ANOVA | Analysis of Variance |
| ATC | Anatomical Therapeutic Chemical |
| AUC <sub>(inf)</sub> | Area under the Plasma Concentration-time Curve from zero hours to |
| AUC <sub>(0-t)</sub> | infinity Area under the Plasma Concentration-time Curve from zero hours to time (t) |
| CBC | Complete Blood Count |
| CFR | Code of Federal Regulations |
| Cmax | Maximum Plasma Concentration |
| CRS | Chronic Rhinosinusitis |
| CRSsNP | Chronic Rhinosinusitis without Nasal Polyposis |
| CRSwNP | Chronic Rhinosinusitis with Nasal Polyposis |
| CT | Computed Tomography |
| DMC | Data Monitoring Committee |
| eCRF | Electronic Case Report Form |
| ECG | Electrocardiogram |
| ECP | Eosinophilic Cationic Protein |
| ELISA | Enzyme-linked Immunosorbent Assay |
| ET | Early Termination |
| EU | European Union |
| FACS | Fluorescence-Activated Cell Sorting |
| FDA | Food and Drug Administration |
| FEF | Forced Expiratory Flow |
| FEV1 | Forced Expiratory Volume in 1 Second |
| FSH | Follicle-Stimulating Hormone |
| FVC | Forced Vital Capacity |

| LIST OF AB | BREVIATIONS |
|---|---|
| GCP | Good Clinical Practice |
| gMean | Geometric Mean |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HIV | Human Immunodeficiency Virus |
| HR | Hazard Ratio |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IgE | Immunoglobulin E |
| IgG4 | Immunoglobulin G4 |
| IEC | Independent Ethics Committee |
| IFN | Interferon |
| IL | Interleukin |
| INS | Intranasal Steroid |
| IRB | Institutional Review Board |
| IXRS | interactive Voice or Web Response System |
| IV | Intravenous(ly) |
| LS | Least-Squares |
| MAb | Monoclonal Antibody |
| MC | Mast Cells |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MPO | Myeloperoxidase |
| PE | Physical Examination |
| PGD2 | Prostaglandin D2 |
| PH | Proportional Hazard |
| PK | Pharmacokinetic(s) |
| PNIF | Peak Nasal Inspiratory Flow |
| RMPA | Replacing Missing Value with Placebo Average |
| SAE | Serious Adverse Event |

| LIST OF ABBREVIATIONS | |
|---|---|
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SF-36 | 36-Item Short Form Health Survey |
| Siglec | Sialic Acid-binding, Immunoglobulin-like Lectin |
| SI Units | International System of Units |
| SNOT-22 | Sino-nasal Outcome Test-22 |
| SOC | System Organ Class |
| t <sub>1/2</sub> | Terminal Elimination Half-life |
| TEAE | Treatment-Emergent Adverse Event |
| TNF | Tumor Necrosis Factor |
| TPS | Total Polyp Score |
| TSLP | Thymic Stromal Lymphopoietin |
| ULN | Upper Limit of Normal |
| UPSIT | University of Pennsylvania Smell Identification Test <sup>TM</sup> |
| VAS | Visual Analogue Scale |
| Vz | Volume of Distribution |
| WBC | White Blood Cell |
| WHO | World Health Organization |

#### **DEFINITIONS**

Adverse Event (AE) An adverse event is any untoward medical occurrence in

a patient or a clinical investigation of subject which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease, whether or

not considered related to the medicinal product.

Intent-to-Treat (ITT)

**Population** 

All randomized subjects

Modified Intent-to-Treat

(MITT) Population

All randomized subjects who take at least one dose of the study drug and have both a baseline and at least one post-

baseline efficacy assessment.

Per-Protocol (PP)

**Population** 

All MITT population subjects who have a week 12 visit

and valid efficacy measurements.

Safety Population All randomized subjects who take at least one dose of

study drug.

Biomarker Population All randomized subjects who has at least 1 sample

obtained for biomarker analysis.

Serious AE (SAE) A serious adverse event (SAE) is an adverse event that

results in any of the following outcomes: death, life-

threatening AE, persistent or significant

disability/incapacity, inpatient hospitalization or prolongation of existing hospitalization, and congenital anomaly/birth defect. A medically significant AE is also

an SAE

Treatment-emergent AE

(TEAE)

AEs with an onset time on or after the time of the initial

dose of study drug or that worsen in intensity or

treatment attribution.

#### 1. INTRODUCTION

#### 1.1 General

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of Allakos, Inc. Protocol AK001-002 [A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Study To Evaluate Multiple Doses of AK001 In Patients With Moderate to Severe Nasal Polyposis]. The purpose of this plan is to provide specific guidelines from which the analysis will proceed. Changes made to the SAP after it has been signed but prior to database lock will be documented in an amendment. Any deviations from these guidelines will be documented in the clinical study report (CSR).

#### 1.2 Protocol Versions

There are four different versions of the protocol governing this document as listed below.

| Version | Country | Comment |
|---|---|---|
| V 1.0 | US | Not applicable |
| V 2.0 | US and Spain | Original used for operation |
| V 2.1 | UK | Primarily, extended the study observation to Week 24 for safety reasons |
| V 2.2 | Netherlands and Belgium | A Biomarker sub-study with optional participation |
| V 2.3 | Germany | Extend the study observation to Week 24; No more than 1 patient wil be randomized every 4 weeks at each site |

As a result of these changes, no implications on the analysis of safety or efficacy is anticipated. However, a section on exploratory analysis of the Biomarkers will be added to the document. The remaining changes in different versions of the amended protocols, mostly impact inclusion and exclusion criteria as well as duration of observation.

#### 2. STUDY OBJECTIVES

## The primary objective is:

To evaluate the effect of each of 2 doses of AK001 separately in combination with an INS versus the INS alone on the reduction in size of nasal polyps as

evaluated by the change from Baseline to Week 12 after the start of treatment in Total Polyp Score (TPS).

## The secondary objectives are:

- 1. To evaluate the effect of each of 2 doses of AK001 separately in combination with an INS versus the INS alone on changes from Baseline to Week 12 after the start of treatment in:
  - a) Size of polyps as evaluated by Lund-Mackay score at selected sites by computed tomography (CT) scan
  - b) Nasal airway patency as evaluated by peak nasal inspiratory flow (PNIF)
  - c) Ability to smell (University of Pennsylvania Smell Identification Test<sup>TM</sup> [UPSIT])
  - d) Patient-reported symptoms of sinusitis (Sino-nasal Outcome Test-22 [SNOT-22] and Visual Analogue Scales [VASs])
  - e) Clinical symptoms improvement scale
  - f) Quality of life (36-Item Short Form Health Survey [SF-36])
- 2. To evaluate the time to first response in TPS
- 3. To evaluate the change in TPS, UPSIT, and patient-reported symptoms of sinusitis over time
- 4. To evaluate the safety and tolerability of each of 2 doses of AK001 separately in combination with an INS during 7 weeks of study drug in patients with moderate to severe nasal polyps and whose symptoms are resistant to INSs

The exploratory objectives (in sites with appropriate capability) are: In all patients, to:

1. Potentially explore markers of Mast Cells (MC) and eosinophils and inflammatory response in blood

In patients with comorbid asthma, to explore the effect of each of 2 doses of AK001 separately in combination with an INS versus the INS alone on changes from Baseline to Week 12 after the start of treatment in:

- 2. TPS
- 3. Pulmonary function (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC], and forced expiratory flow [FEF])
- 4. Asthma-related symptoms (Asthma Control Test<sup>TM</sup> [ACT])
- 5. Use of asthma rescue therapy

## The objective for biomarker analyses is (sub-study; Protocol v2.2):

In patients at slected investigator sites, to evaluate Baseline and post-treatment levels of biomarkers related to the activity of MCs and eosinophils in nasal secretions and blood samples. Evaluations will include change from baseline and effect over time.

#### 3. STUDY DESIGN

This is a Phase 2, randomized, double-blind, placebo-controlled study of the safety and tolerability of AK001 compared with placebo in patients with moderate to severe chronic nasal polyposis and whose symptoms are resistant to treatment with INSs. At least 50% of patients enrolled will have comorbid asthma.

The study will comprise an up to 4-week Screening period and a 4-week run-in period followed by randomization and dosing with AK001 or placebo for 7 weeks followed by a 9-week observation period. There will be 9 scheduled study visits. The total duration of the study will be up to 24 weeks. For UK and Germany, the observation period is extended to 17-week, there will be 10 scheduled study visits. As a result, the total duration of the study for UK and Germany will be up to approximately 32 weeks.

After the Screening period, approximately 70 eligible patients will be enrolled and enter a run-in period of 4 weeks to achieve a stable regimen with a common intranasal topical steroid (NASONEX [mometasone furoate monohydrate] 2 sprays in each nostril twice a day) and discontinue any other intranasal topical steroid. Patients will return to the clinic at the end of the run-in period prior to dosing with study drug for pre-dose evaluations. Patients who continue to meet the eligibility criteria for the study will be randomized, will continue to use NASONEX, and will also receive either 25 mg of AK001 (n=25), 250 mg of AK001 (n=25), or a corresponding placebo (n=20) on Days 0, 21, and 49. The randomization will be stratified based on presence or absence of asthma. Patients will be required to maintain their Baseline treatments for nasal polyposis unchanged throughout participation in this trial.

A Data Monitoring Committee (DMC) will be convened periodically to monitor the safety of patients over the course of the study. Members of the DMC can request the identities of patients' study drugs if needed. Additional information about the DMC can be found in the DMC charter.

A more detailed schedule of events can be found in the protocol Section 4.2. However, the general visit schedule of the study is depicted in the following table.

| | Screening<br>Period | Run-in<br>Period <sup>1</sup> | Treatment Period <sup>2</sup> | | | Post-trea | atment Period | |
|---|---|---|---|---|---|---|---|---|
| Visit | Screening | Run-in | Day 0 | Day 14 | Day 21 | Day 49 | Day 84 | Day 112/ET |
| Day | -56 to -29 | -28 to -1 | 0 | 14±2 | 21±2 | 49±2 | 84±4 | 112±4 or ET |
| Week | [-8 to -4) | [-4 to 0) | 0 | 2 | 3 | 7 | 12 | 16 <sup>3</sup> |

<sup>&</sup>lt;sup>1</sup> The targeted last measurement is day -3, with a visit window of 2 days.

## 4. DETERMINATION OF SAMPLE SIZE

The study will be conducted at approximately 14 investigational sites in the European Union and the United States, and approximately 70 patients will be enrolled.

This study will evaluate the effect of each of 2 doses of AK001 separately in combination with an INS versus the INS plus placebo on the reduction in size of nasal polyps. In an earlier investigational study, the Sponsor observed similar efficacy effect for both the high and low doses administered in this study. Assuming equal efficacy effect of the 2 active treatment arms, a planned sample size of approximately 70 patients (25 mg of AK001 [n=25], 250 mg of AK001 [n=25], and a corresponding placebo (n=20]) will ensure at least 80% power to detect a difference in mean nasal polyp scores between the placebo group (Mean = -0.3; SD  $\leq$ 1.128) and each of the AK001 groups (Mean = -1.9; SD  $\leq$ 2.064) with an alpha of 0.05. PASS 11, Version 11.0.10, was used for this power analysis.

The randomization was enforced with two stratification factors; Region (US vs. non-US), as well as Comorbid Asthma (presence vs. absence). A non-study unblinded statistician assisted with developing the randomization schedule, incorporating it into the IXRS system, and the user acceptance testing (UAT).

<sup>&</sup>lt;sup>2</sup> Measurements could be pre- or post-dose. For complete detail please see protocol section 4.2.

<sup>&</sup>lt;sup>3</sup>24 week for UK and Germany.

The sub-study will be conducted at selected Investigator sites that are participating in the main study. It is expected that approximately 20 patients will participate in the sub-study regarding the biomarker analysis (protocol v2.2).

#### 5. GENERAL ANALYSIS CONSIDERATIONS

The statistical analyses will be reported using summary tables, figures, and data listings. Unless otherwise noted, all statistical testing will be two-sided and will be performed at the 0.05 significance level. Tests will be declared statistically significant if the calculated p-value is < 0.05. Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentage of subjects in corresponding categories.

All summary tables will be presented by treatment group as defined for the population included. Baseline summaries will also include a total summary column pooling across the two groups. Summary tables presenting results by study visit will include all scheduled study visits using informative visit labels (i.e., Baseline, Run-in, Day 0, Week 2, Week 3, Week 7, Week 12 and Week 16/24 or ET – note: Week 16 will be Week 24 for UK and Germany).

Individual subject data obtained from the case report forms (CRFs), central or local clinical laboratories, electrocardiogram (ECG) readers, imaging core laboratories (CT scan), selected IXRS system, and any derived data will be presented by subject in data listings. Listings will include relative study day, where negative values will indicate pretreatment visits, and data collected after discontinuation of study drug will be flagged as follow-up. All data captured on the CRF, including specific descriptions of 'other' and comment fields, will be included on the listings. Listings will be sorted by subject number within each treatment group.

The analyses described in this plan are considered *a priori*, in that they have been defined prior to database lock and prior to breaking the blind. Any analyses performed subsequent to breaking the blind will be considered *post-hoc* and exploratory. *Post-hoc* analyses will be labeled as such on the output and identified in the CSR.

All analyses and tabulations will be performed using SAS® Version 9.4 or higher. Tables, listings, and figures will be presented in RTF format. Upon completion, all SAS® programs will be validated by an independent programmer. In addition, all program output will undergo a senior level statistical review. The validation process will be used to confirm that statistically valid methods have been implemented and that all data manipulations and calculations are accurate. Checks will be made to ensure accuracy,

consistency with this plan, consistency within tables, and consistency between tables and corresponding data listings. Upon completion of validation and quality review procedures, all documentation will be collected and filed by the project statistician or designee.

#### **5.1 Conventions**

The precision of original measurements will be maintained in summaries, when possible. Means, medians and standard deviations will be presented with an increased level of precision; means and medians will be presented to one more decimal place than the raw data, and the standard deviations will be presented to two more decimal places than the raw data.

Summaries of continuous variables that have some values recorded using approximate values (e.g., < or >) will use imputed values. The approximate values will be imputed using the closest exact value for that measurement. For tables where rounding is required, rounding will be done to the nearest round-off unit. For example, if the round-off unit is the ones place (i.e., integers), values  $\ge$  XX.5 will be rounded up to XX+1 while values  $\le$  XX.5 will be rounded down to XX.

For percentages, unless they are calculated to be exactly 0% or 100%, values of very small or very large percentages will be reported as <0.1% and >99.9%.

For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the subjects discontinue due to "lost to follow-up" this reason will be included in the table with a count of 0.

#### **5.2 Standard Calculations**

Variables requiring calculation will be derived using the following formulas:

- **Baseline** A baseline value, unless specified otherwise, is the last non-missing value recorded prior to the first dose of study drug. If an assessment has both a date and time that exactly match the date and time of first dose of study drug, the assessment will be counted as baseline.
- **Study day** For a given date (*date*), study day is calculated as days since the date of first dose of study drug (*firstdose*):

Study day = date – firstdose + 1, where date  $\geq$  firstdose Study day = date – firstdose, where date  $\leq$  firstdose Study day 0 is defined as the day of study drug administration.

- **Days** Durations, expressed in days, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in days = (date2-date1+1).
- Weeks Durations, expressed in weeks, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in weeks = (date2-date1+1)/7.
- **Months** Durations, expressed in months, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in months = (date2-date1+1)/30.4375.
- Years Durations, expressed in years, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in years = (date2-date1+1)/365.25.
- Body Mass Index (BMI) BMI  $(kg/m^2)$  = weight  $(kg) / [[height (cm)/100]^2]$
- Estimated Glomerular Filtration Rate (eGFR) eGFR (mL/min/1.73 m<sup>2</sup>) = 175 × (serum creatinine in mg/dL)<sup>-1.154</sup> × (Age in years)<sup>-0.203</sup> × (0.742 if female) × (1.212 if African American).

Note that age on consent date is collected on the CRF and will not be calculated.

## 5.3 Handling Partial Dates for Adverse Events and Medications

If only a partial date is available and is required for a calculation, the following standards will be applied:

- Start dates
  - a. For missing start day only Day will be imputed as the first day of the month (i.e., 1) with the following exception: if the partial date falls in the same month and year as the date being used in the calculation (e.g., first dose date, informed consent date), then the partial date will be imputed to equal the date being used for the calculation.
  - b. For missing start day and month Day and month will be imputed as the first day of the year (i.e., 1 January) with the following exception: if the partial date falls in the same year as the date being used in the calculation (e.g., first dose date, informed consent date), then the partial date will be imputed to equal the date being used for the calculation.
- Stop dates
  - a. For missing stop day only Day will be imputed as the last day of the month (i.e., 28, 29, 30, or 31)

b. For missing stop day and month - Day and month will be imputed as the last day of the year (i.e., 31 December)

A completely missing start date will be imputed as first dose date of study medication and a completely missing end date will be imputed as study completion date.

The date of last dose of study drug will be taken from the Study Exit Status CRF page whenever available. If this is missing, then the last visit date, excluding the follow-up visit, will be used, unless a blinded data review indicates it was earlier.

Any partial dates will be displayed in data listings without imputation of missing days and/or months (e.g., MAR2016 for missing day, and 2015 for day and month both missing).

#### **5.4 Visit Windows**

Screening period is expected to happen at any time during 56 to 29 days before study Day 0. Upon a successful screening visit, subjects will be enrolled and enter a run-in period of 4 weeks from Day -28 to Day -1 to achieve a stable regimen with a common intranasal topical steroid (NASONEX [mometasone furoate monohydrate] 2 sprays in each nostril twice a day) while discontinuing any other intranasal topical steroid.

Subjects' qualifications will be tested once again before getting randomized into the study on Day 0. Subjects will be expected to be treated for 7 weeks (Day 0 to Day 49), followed by a follow up visits 5 and 9 weeks later (Days 84 and 112). During treatment phase a 2-day margin of error for each visit, and 4-day margin of error for each follow up visit will be acceptable.

However, since study visits do not always take place exactly as scheduled in the protocol, it is necessary to assign the actual observation times to "analysis visit windows" for analysis purposes. Visit windows for each target visit are defined in <u>Appendix A</u>, and will be applied to all (safety, efficacy, etc.) measurements. For each summary and value if there are multiple values within a visit window, the "worst" value as defined in <u>Appendix E</u> will be used for that visit window summary except for all the efficacy endpoints where the rules are described in section 9. These visit windows will be applied to all visits, including scheduled, unscheduled, and early termination visits.

#### 5.5 Review of Blinded Data

A number of analyses may require review of blinded data prior to database lock. The following reviews may occur while the study is ongoing or prior to database lock. Subject ID will be masked in all of these reviews to avoid introducing any bias.

- Concomitant medications are reviewed independent of Subject ID to identify prohibited meds
- ECG data independent of Subject ID.
- Review of adverse event summaries and listings to identify MedDRA preferred terms chosen are consistent with drug's mechanism of action.
- Review of protocol and consent deviations to identify major deviations that would exclude subjects from the per-protocol population.
- Review of subjects with a missing or partial last dose date on the Study Exit Status CRF in order to determine an appropriate imputed date or other missing or partial dates for a parameter of interest; if deemed necessary.
- Reasons for withdrawal which are potentially treatment related

#### 6. ANALYSIS POPULATIONS

The following subject populations will be used for efficacy analyses:

- Intent-to-Treat (ITT) population will include all randomized subjects. Treatment assignment will be based on the randomized treatment.
- Modified Intent-to-Treat (MITT) population will include all randomized subjects
  who take at least one dose of the study drug and have both a baseline and at least
  one post-baseline efficacy assessment, but prior to the 4-week post-dose followup assessment, for at least one of the following efficacy endpoints: TPS, PNIF,
  UPSIT, SNOT-22 or VAS.
- Per-Protocol (PP) population will include all MITT population subjects who have a week 12 visit and valid efficacy measurements. Treatment assignment will be based on the randomized treatment.
- Subjects will be included in their randomized stratum as reflected by the IXRS rather than eCRF.

The Pharmacokinetic (PK) population will include any subject who received study drug and also had a post-dose PK sample drawn, defined as patients with serum concentration data obtained at pre-defined time points.

The Safety population will include all randomized subjects who take at least one dose of study drug. Treatment assignment will be based on the treatment actually received. If a subject receives an incorrect treatment transiently, they will be assigned to the predominant treatment group (i.e., the treatment group for which they received the greater number of doses).

Biomarker analyses will be performed in the Biomarker Population, defined as patients with at least 1 sample obtained for biomarker analysis.

Should there be a for-cause reason to disqualify data from any non-compliant site, a Note-To-File letter, signed by the Sponsor, will be provided to InClin Biostatistics to do so. This Note-To-File letter should include description of the event/reason and an unbiased assessment of impact. A subset of the analyses will be run with and without this data to further assess the impact.

#### 7. STUDY POPULATION

## 7.1 Subject Disposition

Subject disposition information will be summarized for all subjects by treatment group, overall and by region, country and site. Summaries will include: the number of randomized subjects, the number of subjects in each analysis population, the number of subjects completing the study (and subsets completing the study on and off treatment), all reasons for discontinuation of study drug and study, and the primary reason for discontinuation of study.

The visit schedules and their timing are given in the table in Section 3 as given in Section 4.2 of the protocol:

A listing of all early discontinuations from study drug, as well as discontinuation from the study will be provided.

#### 7.2 Protocol Deviations

In accordance with ICH E3, Sponsor-defined eligibility violations and post-randomization protocol deviations will be identified and listed separately by study site and subject. Sources for these deviations may include IXRS, Trial Management or the clinical database. Deviations will be classified as follows (also see Appendix G):

Deviation type/code as provided by Sponsor includes but is not limited to the following:

- Informed consent.
- Randomization error
- Safety
- Efficacy
- IP / Treatment deviation
- Other protocol deviations

Deviations are then categorized into:

- Major
- Minor

A listing and tabulation of protocol deviations will be provided.

## 7.3 Demographic and Baseline Characteristics

Demographic variables to be summarized include the following: age at informed consent, gender, ethnicity, race, geographic region, height, weight, and body mass index (BMI). Height (in cm) and weight (in kg) will be measured at Screening, and BMI will be calculated. Weight will also be measured on Days 0 and 112 or ET.

Demographic and baseline characteristics will be summarized for all the analysis populations (ITT, MITT, and Safety). Summaries will also be provided by region (US and non-US), for the MITT population.

#### 7.4 Medical History

Verbatim terms on case report forms will be mapped to preferred terms and system organ classes using the Medical Dictionary for Regulatory Activities (MedDRA) (version 16.0 or higher).

The number and percentage of subjects with a given medical and/or surgical history will be summarized for each system organ class. Summaries will be provided for the Safety population. The verbatim and coded medical histories will be included in a listing.

#### 7.5 Physical Examinations

A complete PE will be performed by either the Principal Investigator or a qualified Subinvestigator at Screening. A complete PE will include the following body system or

organ assessments: skin; head, eyes, ears, nose, and throat (HEENT); thyroid; lungs; cardiovascular system; abdomen; extremities; lymph nodes; and a brief neurological examination. Clinically significant findings will be documented.

A symptom-directed PE, including assessments of possible infusion site reactions, will be performed by either the Investigator or a qualified Subinvestigator pre-dose on Days 0, 21, and 49; and on pre- or post-dose on Days 14, 84 and 112 or ET. New abnormal PE or worsened findings will be documented by the Investigator or qualified Subinvestigator at the next scheduled visit. Whether physical exam was performed, along with body system and any clinically significant findings will be summarized by visit, and a detailed listing will be provided.

Symptom directed physical exams will tabulate injection site reactions, corresponding AE if any, and whether it was worsened or rise to levels of clinically significant outcome.

Physical and neurological examination results will be presented in by-subject listings. The results of complete physical and neurological examinations performed at screening will be summarized by body system. Evaluations based on the targeted examinations performed at subsequent visits will be summarized in a treatment-emergent fashion. For the physical examination, each body system is assessed as Normal or Abnormal, and if Abnormal, then Clinically Significant or Not Clinically Significant. For the neurological examination, each body system is assessed as Normal or Abnormal, and if Abnormal, then Clinically Significant or Not Clinically Significant.

Summaries will present the number and percentage of subjects within each category by visit and by body system/parameter evaluated.

#### 7.6 Vital Signs

Body temperature, supine systolic and diastolic blood pressure, pulse, and respiratory rate will be measured at Screening and on Days -3, 0, 14, 21, 49, 84, and 112 or at ET. On Days 0, 21, and 49, vital signs will be measured pre-dose, and every 15 minutes after the start of infusion, as well as immediately following the end of infusion. All vital signs will be measured after the patient has been in the supine position for ≥5 minutes. These measurements include systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature.

## **7.7 ECG**

12-Lead ECG will be collected only at screening between Days -56 to -29. Mean heart rate, RR, PR, QRS, QTcB and QTcF along with abnormalities will be summarized and a listing will provide more detailed by-subject data.

#### 7.8 Fecal Collection

Fecal samples will be collected at Screening for ova and parasite tests.

#### 7.9 Adverse Events

Information regarding AEs will be obtained from the time of the first study drug administration until completion of the last study-related procedure (Day 112 or ET). Information regarding serious adverse events (SAEs) will be obtained from the time the patient signs an ICF until completion of the last study-related procedure (Day 112 or ET). Duration (start and stop dates and times), severity, outcome, treatment, and relation to study drug will be recorded on the eCRF.

#### 7.10 Laboratory Values

Serum pregnancy (at Screening and Days -3, 21, 49 and 112 or ET), hematology and chemistry (at Screening, Days -3, 14, 21, 49, 84, and 112 or ET), and urinalysis (at Screening, Days -3, 14, 49, 84, and 112 or ET) laboratory results will be collected, listed by subject and visit, and tabulated by visit for each parameter.

## 7.11 Anti-Drug Antibody (ADA)

Blood will be collected for determination of ADA pre-dose on Day 0 and, should a related AE suspected of being associated with immunogenicity occur, post-dose, as well as on Day 112 or ET. Should these results be available at the time of developing the TLFs, a summary and listing will be provided.

## 7.12 Prior and Concomitant Medications

Verbatim terms on case report forms will be mapped to Anatomical Therapeutic Chemical (ATC) class and Generic Drug Names using the World Health Organization (WHO) dictionary (WHODDE B2, March 1, 2015 release or higher).

Prior and concomitant medications include both prescribed and over-the-counter medications. Prior medications are those medications started within the 30 days before Screening. Concomitant medications are those medications taken at the start of study drug or initiated after the initial dose of study drug. Prior medications and concomitant medications will be summarized separately for each treatment by WHO ATC level 1

term, ATC level 3 term and Preferred Term (generic name) with frequency and percentage of subjects in each dosing arm using each prior medication and each concomitant medication. At each level of subject summarization, a subject is counted once if he/she reported one or more medications at that level. Each summary will be ordered alphabetically by each level of ATC class and generic drug name within each level of ATC class. Prior and Concomitant medications will also be listed separately with these elements as well as the verbatim drug name.

The overall summary and subsets of concomitant medications will be provided for all the analysis populations. The summary of prior medications will be provided only for the Safety Population.

#### 8. EFFICACY ANALYSES

The primary efficacy analysis will be based on the MITT population. Additional supportive efficacy analyses will be performed using the PP population. Selected sensitivity analyses will be performed using the ITT population.

## 8.1 Efficacy Variables

## 8.1.1 Primary Efficacy Variable

The primary endpoint of this study is the reduction in TPS values from Baseline to Week 12 after the start of treatment. Polyps will be evaluated in each nostril by means of nasal endoscopy and graded based on polyp size, resulting in scores of 0 to 4 as indicated in <a href="Appendix F">Appendix F</a>. The TPS is the sum of the left and right nostril scores. The TPS values for efficacy analyses will be determined from blinded central evaluations of nasal endoscopies performed at Screening, on Day -3, pre-dose on Days 21 and 49, and on Days 84 and 112 or ET. Videos of the endoscopies will be evaluated by independent blinded reviewer.

## 8.1.2 Secondary Efficacy Variables

The following secondary clinical endpoints will be evaluated from Baseline to Week 12 after the start of treatment on changes in:

- Size of polyps as evaluated by Lund-Mackay score (in <u>Appendix F</u>) at selected Investigator sites by CT scan on Days -3 and 84 or ET
- Nasal airway patency as evaluated by PNIF pre-dose on Days 0 and 21 and on Days 84 and 112 or ET

- Ability to smell by UPSIT (in <u>Appendix F</u>) pre-dose on Days 0, 21, and 49 and on Days 14, 84, and 112 or ET
- Patient-reported symptoms of sinusitis by SNOT-22 (in <u>Appendix F</u>) pre-dose on Days 0, 21, and 49, and on Days 14, 84, and 112 or ET and VASs on Day -3, pre-dose on Days 0, 21, and 49; and on Days 14, 84, and 112 or ET
- Clinical symptoms improvement scale (in <u>Appendix F</u>) on Day -3, pre-dose on Days 0, 21, and 49; and on Days 14, 84, and 112 or ET
- Quality of life by SF-36 (in <u>Appendix F</u>) pre-dose on Days 0, 21, and 49 and on Days 84 and 112 or ET

The secondary efficacy variables also include the following:

- Time to first response in TPS
- Change in TPS, UPSIT, and patient-reported symptoms of sinusitis over time
- Safety and tolerability of each of 2 doses of AK001 separately in combination with an INS

## 8.1.3 Exploratory Efficacy Variables

Several exploratory analyses are pre-specified (additional *post hoc* analyses may be performed):

In all patients, to

 Potentially explore markers of MCs and eosinophils and inflammatory response in blood

In patients with comorbid asthma, to explore the effect of each of 2 doses of AK001 separately in combination with an INS versus the INS alone on changes from Baseline to Week 12 after the start of treatment in:

- TPS
- Pulmonary function (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC], and forced expiratory flow [FEF]) assessed using spirometry (from Baseline to Week 7)
- Asthma-related symptoms (Asthma Control Test<sup>TM</sup> [ACT]) in <u>Appendix F</u>
- Use of asthma rescue therapy

#### **8.2 Adjustments for Covariates**

The models for analyses of the primary endpoint (change in TPS) will include the treatment group, time, interaction between treatment group and time.

Also, all analyses will include presence or absence of asthma as the only stratification variable in the model.

## 8.3 Handling of Dropouts or Missing Data

The occurrence of missing data could potentially lead to bias and misleading conclusions. Therefore, strenuous efforts and plans are in place to obtain all scheduled efficacy assessments from all randomized subjects, regardless of whether or not they remain on study treatment. In addition, multiple sensitivity analyses will be performed to examine robustness of the results of the pre-specified primary analyses. These sensitivity analyses will be described in greater detail in later sections of this document.

## 8.4 Interim Analysis and Data Monitoring

No interim analyses are planned for evaluating efficacy. However interim safety monitoring will be performed according to the DMC charter.

#### 8.5 Examination of Subgroups

Subgroup analyses are to be performed for the primary and the exploratory efficacy variables with subjects categorized by the presence of asthma. If adequate data is available, gender (male, female), and age (<median, ≥median) will be used as covariates as well.

## 8.6 Multiple Comparisons/Multiplicity

Each active treatment group will be compared separately with the placebo group by utilizing a mixed effect repeated measures analysis of variance (ANOVA) model with specific contrast statement for Week 12 as well as other time points for each comparison separately. Adjustment in alpha for multiple comparisons will be controlled according to the Hochberg method, in which, if the efficacy comparison of the high active arm versus placebo is statistically significant at the 0.05 level, no penalty will be assessed to the comparison of low active arm versus placebo. Otherwise, the low active arm versus placebo will be compared at the 0.025 level.

#### 8.7 Multicenter Studies

The study will be conducted at approximately 14 investigational sites in the European Union and the United States, and approximately 70 patients will be enrolled.

Because the study will include a large number of study sites, relative to the total number of subjects, the effect of study site will not be included in the statistical analysis models. However if a highly influential site is identified, the differences between treatment groups will be examined with and without the influential site.

#### 9. METHODS OF EFFICACY ANALYSIS

For all efficacy analyses, if there are multiple values within a visit window, the ontreatment value whose date is closest to the scheduled date shall be used for the summary. In the case that more than one on-treatment value is equidistant from the scheduled date, the later will be used

#### 9.1 Primary Efficacy Analyses

There are therefore three primary null hypotheses to consider:

 $H_01$ : There is no difference between AK001 (250 mg or 25 mg) in combination with NASONEX and NASONEX alone in reduction in size of nasal polyps as evaluated by the change from Baseline to Week 12 in TPS

 $H_02$ : There is no difference between AK001 250 mg (high dose) in combination with NASONEX and NASONEX alone in reduction in size of nasal polyps as evaluated by the change from Baseline to Week 12 in TPS

H<sub>0</sub>3: There is no difference between AK001 25 mg (low dose) in combination with NASONEX and NASONEX alone in reduction in size of nasal polyps as evaluated by the change from Baseline to Week 12 in TPS

The primary analyses will be based on the MITT population, defined as all subjects randomized who receive at least 1 dose of study drug and have a valid Baseline measurement and at least 1 post-baseline efficacy assessment. Subjects will be analyzed for efficacy according to the group to which they were randomized.

The primary analysis specification refers to "number of subjects retained at week 12" where "number of subjects retained at visit X" is defined as follows: If a subject has an on-treatment assessment with a non-missing score for any of efficacy measurements at visit X, or at any scheduled visit subsequent to X, then this subject is defined to be

retained at visit X. Otherwise the subject is defined to be not retained at visit X. Note that this is a per-subject definition, not a per-endpoint definition.

The effect of each of 2 doses of AK001 separately in combination with an INS versus the INS alone on the reduction in size of nasal polyps as evaluated by the change from Baseline to Week 12 after the start of treatment in TPS will be displayed for each treatment group by study visit using summary statistics, including the number of observations, the mean, median, standard deviation (SD), and range (min, max). Each active treatment group will be compared separately with the placebo group for change from Baseline in TPS by using a mixed effect repeated measures analysis of variance (ANOVA) model with specific contrast statement for Week 12 and for each comparison separately. Adjustment in alpha for multiple comparisons will be controlled according to the Hochberg method, in which, if the efficacy comparison of the high active arm versus placebo is statistically significant at the 0.05 level, no penalty will be assessed to the comparison of the low active arm versus the placebo arm. Otherwise, the low active arm versus the placebo arm will be compared at the 0.025 level.

The dependent variable will be the change from baseline in TPS (blinded centralized nasal endoscopy score) at Week 12. The mixed model, as the primary analysis of the primary endpoint, will include fixed effects for treatment group (three levels), asthma (two levels: presence versus absence), and baseline TPS score. The Kenward and Roger method of calculating the denominator degrees of freedom will be used for the tests of fixed effects. Treatment comparisons to placebo will be established using contrast statements at Week 12.

#### 9.2 Sensitivity Efficacy Analyses of Primary Endpoints

## 9.2.1 Analysis for TPS in Presence of Missing Data

Because the occurrence of missing data could potentially lead to bias, strenuous efforts will be made to obtain all scheduled efficacy assessments from all randomized subjects, regardless of whether or not they remain on study treatment.

Missing values will be imputed by replacing the missing value with the average value of the placebo group at the specific time point

At the conclusion of imputation of the missing data, the same identical analysis as described for the primary endpoint (Section 9.1) will be once again conducted to examine the robustness of the outcome.

## 9.2.2 The Analysis with TPS including Time as a Repeated Factor

The dependent variable will be the change from baseline in TPS (blinded centralized nasal endoscopy score) at Week 12. The mixed model, as the primary analysis of the primary endpoint, will include fixed effects for treatment group (three levels), asthma (two levels: presence versus absence), time (weeks 0, 3, 7, 12, and 16[ET]) in which case, baseline TPS and subject as random effects (using SAS Repeated statement), and the interaction between treatment effect and time may be included in the model. The Kenward and Roger method of calculating the denominator degrees of freedom will be used for the tests of fixed effects. Treatment comparisons to placebo will be established using contrast statements at Weeks 2, 3, 7, 12 and 16.

## 9.2.3 Analysis of TPS in Absolute Value and Percent Change from Baseline

Additional efficacy measures will be analyzed in support of the primary efficacy endpoint results. In addition to change from Baseline in TPS, absolute values and percentage changes from Baseline will be analyzed separately using the same repeated measures model described above (Section 9.2.2).

## 9.2.4 Alternate Analysis Population

The primary efficacy analyses of TPS will be repeated using the ITT and Per Protocol population based on similar models described in Sections 9.1 and 9.2.2.

## 9.2.5 Time to Response

Time to response will be compared between all 3 treatment groups by summarizing number and number (%) of subjects with response, Mean, Standard Deviation, Range, and Median time to response for those with response. In addition, time to response will be analyzed using Kaplan-Meier curve supplemented by the Cox Proportional hazard model to estimate both the median and HR comparing across the groups.

Response will be defined for each of the following endpoints: TPS, PNIF, UPSIT, SNOT22, and VAS as 50% reduction from baseline. For TPS only, responders will be also defined as those with 1-point reduction from baseline. Kaplan-Meier method and Cox PH model will be utilized to analyze time to first response. The 25<sup>th</sup>, 50<sup>th</sup> (Median) and 75<sup>th</sup> percentiles will be provided by treatment/dose group along with "survival" curves, 95% confidence interval and log-rank test p-value. In addition, HR, its 95% confidence interval and the associated p-value will be also presented.

## 9.2.6 Subgroup Analyses

Subgroup analyses are to be performed for the primary efficacy variable using repeated measures analysis of variance for the following subgroups:

- Comorbid asthma (to be defined on the presence or absence of asthma)
  - Yes
  - o No
- Age
  - < Median
  - $\circ \geq Median$
- Gender
  - o Male
  - o Female
- Response (responders are defined as subjects with 50% or 1-point reduction in total TPS score)
  - Yes
  - o No

#### 9.3 Secondary Efficacy Analyses

The primary population for secondary efficacy analyses will be the MITT population.

- Size of polyps, as evaluated by Lund-Mackay score at selected Investigator sites by CT scan (CT scans are optional and will only be done at Investigator sites at which appropriate and timely regulatory approval or authorization can be granted) (Appendix F) will be measured for six different components of the system, each with possible score of 0=absence; 1=partial opacification; and 2=complete opacification with a total score of 0 to12. Descriptive statistics will be provided by treatment groups for each component of the system and the total score. Change from baseline in total score will be compared between each of the high and low dose AK001 and Placebo using an ANOVA model.
- Change from baseline in PNIF will be compared across the groups using a similar repeated measure ANOVA as described before. Contrast statements will be built to highlight differences at Weeks 3, 12 and 16.

- UPSIT (<u>Appendix F</u>): Descriptive statistics of scoring correct answers (Out of 40 possible correct answers) will be provided by treatment groups. Should it be feasible, score for each odorant will be listed along with the total score. The UPSIT total score will be compared between the groups using a repeated measure ANOVA with contrast statements for comparison at week 12 as well as other time points in the study. It is expected that each subject will respond to each of the Odorants. Missing data will be assumed to be a wrong response and no imputation will be performed to replace.
- Patient-reported SNOT-22 (<u>Appendix F</u>): Five most important items will be listed and summarized for each treatment group. Change from baseline in total score of the five most important items, as well as all items, will be compared between the treatment groups over time using repeated measure ANOVA described before. Contrast statements will be included to compare high and low dose AK001 to placebo at different visits. The missing answers will be imputed by average score of the items present. In other words, missing values will be imputed by the total score divided by the total number of non-missing items with value.
- VAS scale of 0-10 (<u>Appendix F</u>): For each of the five symptoms of rhinosinusitus (Anterior nasal discharge, Posterior nasal discharge, Nasal congestion, blockade, or obstruction, Decreased sense of smell, and Facial pain or pressure), VAS scores will be categorized into mild (0,1,2), moderate (3,4,5,6), and severe (7,8,9,10). Number (%) of subjects in each category will be summarized by treatment group. Change from baseline (Week 0) to each visit for each VAS score from different symptoms will be computed and compared across the treatment groups using a repeated measure ANOVA with contrast statements as described before. Change from baseline in individual symptoms as well as the total VAS score across all symptoms will be analyzed similarly. Missing VAS score will be imputed by average of the non-missing values.
- Clinical symptoms improvement scale (<u>Appendix F</u>): Change from baseline in VAS (0-10) Clinical Symptoms Improvement Scale will be compared over time across the treatment groups using a repeated measures ANOVA model with contrast statements at each visit.
- SF-36 (Appendix F): Change from baseline in total SF-36 score will be compared over time across the treatment groups using a repeated measures ANOVA model with contrast statements at each visit. Missing item values will be imputed by the average score of the category that the question belongs to. These categories are groups of questions with 3, 5 and 6 possible responses as indicated in Appendix F.

## 9.4 Exploratory Efficacy Analyses

Markers of MCs and eosinophils and inflammatory response in blood will be summarized descriptively by mean, median, standard deviation, min and max across groups.

In the subgroup of patients with comorbid asthma, the following analyses will be conducted:

- Use of asthma rescue therapy summarized by number and percentage. Change from baseline to Week 12 will be displayed using a shift table. Scoring the rescue medication question ACT4 by 4, 3, 2, 1, and 0 to perform change from baseline comparison between groups
- Change from screening in pulmonary function as evaluated by FEV1, FVC, and FEF (could be expiratory volume or percentage of lung capacity) will be compared across treatment groups using the same repeated measures ANOVA model described earlier.
- Change from baseline in total ACT score will be compared over time across the treatment groups using a repeated measures ANOVA model with contrast statements at each visit. The missing answers will be imputed by average score of the non-missing values as described earlier.

## 9.5 Pharmacokinetic And Biomarker Analyses

A listing of concentration data and time of sample collection relative to dosing will be generated. Pharmacokinetic parameters will be estimated using non-compartmental methods and compared across the groups using an ANOVA model. Baseline covariates may be added to the model as needed.

At selected investigator sites, biomarkers related to eosinophilic and mast cell (MC) inflammation will be evaluated in nasal secretions and blood samples collected at Days - 3, 14, 21, 49, and 112 or Early Termination (ET) from patients who consent to participate in the analysis. For each biomarker (ECP, histamine, tryptase, prostaglandins, leukotrienes, chymase, carboxypeptidase A3, cytokines, chemokines, and growth factors), the following analyses will be performed:

• Changes from Baseline to Week 16 after the start of treatment:

The effect of 2 different dose levels of AK001 separately in combination with INS versus the INS alone on each of biomarkers as evaluated by change and percent change from baseline to Week 12 after the start of treatment will be displayed for each treatment group by study visit using summary statistics, including the number of observations, the mean, median, standard deviation (SD), and range (min, max). The AK001 25 mg and 250 mg subjects will be compared to placebo according to a mixed effect repeated model which will include treatment, stratification factor (comorbid asthma; if feasible), and baseline as covariates. Each active treatment group will be compared separately with the placebo group for change and percent change from baseline using a similar model if data permits.

#### • Effects over time:

The change and percent change from baseline over time for AK001 25 mg and 250 mg subjects will be compared to placebo according to a repeated measured mixed effect model which will include treatment, stratification factor (comorbid asthma; if feasible), time (weeks 2, 3, 7, and 16[ET]), baseline, and the interaction (if feasible) between treatment and time. Treatment comparisons to placebo will be established using contrast statements at Weeks 2, 3, 7, and 16. If adequate data exists, the same analysis will be repeated to compare each AK001 dose level to placebo. The estimated LS mean and standard error of change and percentage changes from Baseline over time will be plotted.

#### 10. SAFETY ANALYSES

All safety analyses will be based on the Safety population.

Safety and tolerability will be assessed throughout the study by monitoring and evaluating TEAEs, including any complications resulting from the IV infusion, and changes in vital signs and in clinical safety laboratory test (including ADA) and PE findings. All safety and tolerability endpoints will be summarized by treatment. Baseline for all safety endpoints will be defined as the last recorded observation before the administration of the IV infusion of study drug. Safety measures, including AEs, clinical safety laboratory tests (including ADA), vital signs, PEs, and concomitant medication usage, will be summarized descriptively. For quantitative variables, descriptive statistics, including number of observations, means, medians, SDs, and ranges, will be provided for the values themselves as well as for the changes from Baseline by treatment group at

each study visit. Qualitative variables will be summarized using counts and percentages in each treatment group at each study visit.

#### **10.1 Adverse Events**

Adverse events will be coded to System Organ Class (SOC) and preferred term using MedDRA (version 16.0). The coding process is described in the Data Management Plan.

The tabular summaries will be provided for AEs, with the number and percentage of subjects reporting each type of event presented by each treatment group and placebo. If a subject reports the same preferred term more than once, it is counted only once within that category. Further, for a given tabulation, the preferred term will only be counted once at its worst severity and strongest relationship to treatment.

Adverse events will be regarded as treatment-emergent (TEAE) if they start on or after the time of first dose of study drug administration or if they were present prior to the first dose of study drug administration and increased in severity or relationship to study drug while on study drug.

The following summaries for <u>TEAEs</u> will be provided:

- An overall summary table of TEAEs by SOC and preferred term.
- Subject incidence of TEAEs by maximum severity, SOC, and preferred term.
- Subject incidence of TEAEs by MedDRA SOC, preferred term, and strongest relationship to study drug (Related/Not Related). Events reported as "Possibly Related," or "Related" will be included in the Related category. Events reported as "Unlikely Related" or "Not Related" will be included in the Not Related category. At each level of subject summarization a subject is classified according to the strongest relationship, as determined by the investigator, if the subject reported one or more events. AEs with a missing relationship will be considered related for this summary.
- Subject incidence of TEAEs leading to withdrawal by SOC and preferred term.
- Subject incidence of serious TEAEs (SAEs) by SOC and preferred term

All AEs will be collected starting from the first study drug administration through Day 112 or ET. Severity will be assessed by the Investigator using the protocol-defined grading scales (Section 11.1). All AEs will also be judged by the Investigator as to whether they are clinically significant and related to study drug.

<u>Post-treatment AEs</u> are defined as the subset of TEAEs that have an onset more than 7 days after the last dose of study drug or that worsen in intensity or treatment attribution. A summary of post-treatment adverse events by MedDRA system organ class and preferred term will be provided along with a flag in the overall listing.

Summaries for subsets of TEAEs of interest (Allakos AE Groupings) and planned subgroup analyses (e.g., by demographics) are described in the sections following.

All AEs will be presented in a data listing. In addition, listings will also be provided for SAEs (including subsets for fatal and non-fatal SAEs), AEs leading to dose reduction and/or interruption, AEs leading to discontinuation of study drug, and AESIs.

#### 10.1.1 Selected Subsets of Adverse Events

There are no known adverse events of special interest. Should any be noted during the study, they will be flaged in the listings.

## 10.1.2 Subgroup Analyses

The summaries of Allakos AE groupings described in Section 10.1.1, as well as the most common TEAEs (occurring in more than 20% in any treatment group), will be repeated for the following subgroups of subjects:

- Asthma: presence/absence
- Age group: < median and ≥ median
- Gender: male/female

Other subgroup analyses of interest may be identified during data review (e.g., based on concomitant medications or medical conditions).

#### 10.2 Clinical Laboratory Evaluation

Safety laboratory tests include serum chemistry, hematology, urinalysis and ADA findings.

Central laboratory data are transferred electronically by Covance. The Data Transfer Specification document provides a detailed description of the content and format of the laboratory datasets. Both conventional units and International System of Units (SI) are provided and will be summarized in separate tables and listings. The eGFR values will be calculated using the formula provided in Section 5.2 and will be included in the tables and listings for clinical chemistry parameters. Results from local laboratories are entered

into the CRF by the site; these will not be included in summary tabulations but will be included in the data listings together with the corresponding normal ranges. Values for local laboratory parameters will be converted to the corresponding alternative units, either conventional or SI, depending on how reported.

For the summary tabulations of laboratory results, Baseline is defined as the last non-missing value prior to first dose of study drug. Laboratory tests obtained on the date of the first dose will be assigned to pre-treatment; the relative times of blood sampling and dosing will be checked programmatically to confirm this assumption. For each analyte, Baseline values will be restricted to those subjects in the safety population for whom there is at least one post-Baseline value (either overall or for the corresponding target visit).

Visit windows are used when results are presented by target visit (see <u>Appendix A</u>). For each analyte, if a subject has multiple values within a visit window, the "worst" value as defined in <u>Appendix E</u> will be used for that visit window summary.

Descriptive statistics will be used to summarize continuous laboratory results at Baseline, each post-baseline visit, and the change from Baseline for each visit; the last available on-treatment value will also be summarized. For each visit, changes from baseline will also be summarized by n (%), Mean, Median, SD and (Min, Max) for continuous laboratory parameters. In addition, continuous laboratory parameters will be summarized by shift table according to changes from Baseline relative to the reference range (low, normal, high) at Baseline and each post-baseline time point. Missing n (%) will be indicated in all tables

Categorical laboratory parameters will be summarized by treatment group for each target visit using counts and percent of subjects in each category. A shift table will also be presented for categorical parameters. Missing categories will be included in the shift tables.

Thresholds for potentially clinically significant (PCS) laboratory abnormalities are defined in <u>Appendix B</u> for selected parameters. When there are thresholds provided for low and high values, they will be handled separately. Summaries will include the number and percent of subjects with treatment-emergent PCS values, restricted to those subjects in whom the values represent a post-Baseline worsening (PCST); the number meeting criteria at Baseline will also be summarized. A PCST is defined as any PCS event that happened at any post-Baseline visit and has a value more out of range than the value for a particular test at Baseline (see <u>Appendix E</u> for directionality of worsening).

Listings of laboratory parameter results will be presented. Listings will include all laboratory flags provided by the central laboratory in the data transfer as well as flags for those that meet criteria for being PCS (whether or not a treatment-emergent worsening); additionally, results evaluated by the investigator as abnormal/clinically significant will be flagged in the listing.

Separate listings for each hematology, chemistry, and urinalysis parameter will include only subjects with treatment-emergent PCS values and, for these subjects, all laboratory results for the parameter meeting PCS criteria and related parameters (e.g., ALT, AST, bilirubin, neutrophils, WBC, etc.) will be provided.

#### 10.3 Vital Signs

For the summary tabulations of diastolic blood pressure, systolic blood pressure, pulse rate, temperature, and respiratory rate at baseline, baseline will be defined as the last non-missing value prior to the first dose of study drug. Pre-dose and post-dose (target 2 hours post-dose for seated and standing blood pressure and pulse and hourly for at least 4 hours for temperature and respiratory rate) in each parameter will be summarized using descriptive statistics. Change from baseline in these vital signs will also be calculated and summarized.

Vital sign measurements subsequent to Day 0 will be summarized descriptively by target visit using the visit windows defined in <u>Appendix A</u> and the last available on-treatment visit; These include seated blood pressure and pulse, temperature, respiratory rate, and body weight. If a subject has multiple values within a visit window, the "worst" value as defined in <u>Appendix E</u> will be used for that visit window summary.

Potentially clinically significant vital sign changes are defined for selected parameters in Appendix C. When there are thresholds provided for low and high values, they will be handled separately. Summaries will include the number and percent of subjects with treatment-emergent PCS values, restricted to those subjects in whom the values represent a post-Baseline worsening (PCST). A PCST is defined as any PCS event that happened at any post-Baseline visit and has a value more out of range than the value for a particular parameter at Baseline (see Appendix E for directionality of worsening).

Listings of vital sign measurements including height at Screening will be presented. Listings will flag results that meet criteria as being PCS (whether or not a treatment emergent worsening).
Separate listings for each vital sign parameter will include only subjects with treatmentemergent PCS values and, for these patients, all corresponding vital sign results will be provided.

#### 10.4 Prior and Concomitant Medications

Prior and concomitant medications will be summarized by ATC Class 1, ATC Class 3, and preferred term throughout the whole study.

#### 11. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

Changes made to the SAP after it has been signed but prior to database lock will be documented in an amendment. Any important changes made to the analysis and required in response to data review, will be described in the Clinical Study Report (CSR).

#### 12. REFERENCES

- 1. Hedman J, Kaprio J, Poussa T, Nieminen MM. Prevalence of asthma, aspirin intolerance, nasal polyposis and chronic obstructive pulmonary disease in a population-based study. Int J Epidemiol 1999;28(4):717-22.
- 2. Mygind N, Dahl R, Bachert C. Nasal polyposis, eosinophil dominated inflammation, and allergy. Thorax 2000;55 Suppl 2:S79-83.
- 3. Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, et al. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl 2012(23):3 p preceding table of contents, 1-298.
- 4. Pearlman AN, Chandra RK, Conley DB, Kern RC. Epidemiology of nasal polyps. In: Nasal Polyposis, eds. T.M. Onerci and B.J. Ferguson. Springer-Verlag: Berlin Heidelberg 2010. In.
- 5. Bachert C, Gevaert P, Holtappels G, Johansson SG, van Cauwenberge P. Total and specific IgE in nasal polyps is related to local eosinophilic inflammation. J Allergy Clin Immunol 2001;107(4):607-14.
- 6. Kiwamoto T, Kawasaki N, Paulson JC, Bochner BS. Siglec-8 as a drugable target to treat eosinophil and mast cell-associated conditions. Pharmacol Ther 2012;135(3):327-36.
- US Department of Health and Human Services. Common Terminology Criteria for Adverse Events Version 4.0. 28May2009. Available from: http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE\_4.03\_2010-06-14\_QuickReference\_8.5x11.pdf. Accessed 01Feb2016.

#### **APPENDICES**

#### Appendix A: Visit Windows

The visit windows do not apply to the follow-up visits, which are always assigned as follow-up, regardless of when they occur. Unscheduled and early termination visits are included in the windowing algorithm.

Visit windows for efficacy assessments are defined in the following table. In case of multiple values, the one closest to the intended collection time will be chosen.

| Window Label | Time Interval (Study Day <sup>[1]</sup> ) | Scheduled Day |
|---|---|---|
| Screening | -56 to -29 | -42 |
| Run-in | -28 to -1 | -14 |
| Day 0 Predose | 0 | 0 |
| TP: Day 0 | 0 to 3 | 0 |
| TP: Week 2 | 4 to 17 | 14 |
| TP: Week 3 | 18 to 35 | 21 |
| TP: Week 7 | 36 to 63 | 49 |
| FU: Week 12 | 64 to 98 | 84 |
| FU: Week 16 | ≥99 | 112 |
| FU: Week 24 <sup>[2]</sup> | Not Applicable to efficacy | Not Applicable to efficacy |

<sup>[1]</sup> Calculated as in Section 5.2.

<sup>[2]</sup> Week 24 applies to safety data in UK and Germany only, with no impact on efficacy.

Appendix B: Criteria for Determining Potentially Clinically Significant Values in Laboratory Test Results

| Test | Criteria - System | Criteria – |
|---|---|---|
| | International Units | <b>Conventional Units</b> |
| Hemoglobin | Female: $\leq$ 95 g/L; | Female: $\leq 9.5 \text{ g/dL}$ ; |
| | Male: $\leq 115 \text{ g/L}$ ; | Male: $\leq 11.5 \text{ g/dL}$ ; |
| | Decrease of $\geq 20\%$ | Decrease of $\geq 20\%$ |
| Hematocrit | Female: $\leq$ 0.32; Male: $\leq$ | Female: ≤ 32%; |
| | 0.37 | Male: ≤ 37% |
| WBC count | $\leq 2.8 \times 10^9 / L$ | $\leq 2800/\mu L$ or $\geq$ |
| | $\geq 16 \times 10^9/L$ | 1600/μL |
| Neutrophils | $\leq 1.0 \times 10^9 / L$ | $\leq 1000/\mu L$ |
| Eosinophils | $\geq 0.7 \times 10^9/L$ | $\geq 700/\mu L$ |
| Platelet count | $\leq 75 \times 10^9/L$ | $\leq 75 \times 10^3/\mu L$ |
| | $\geq 700 \times 10^9 / L$ | $\geq 700 \times 10^3/\mu L$ |
| Sodium | <130 mmol/L | <130 mEq/L |
| | >150 mmol/L | >150 mEq/L |
| Potassium | < 3.0 mmol/L | < 3.0 mEq/L |
| | > 5.5 mmol/L | > 5.5 mEq/L |
| Calcium | < 1.75 mmol/L | < 7.00 mg/dL |
| | > 3.00 mmol/L | > 12.00 mg/dL |
| Triglycerides, | > 3.39 mmol/L | > 300 mg/dL |
| fasting/nonfasting/unknown | | |
| Glucose, | < 2.775 mmol/L | < 50 mg/dL |
| fasting/nonfasting/unknown | >13.875 mmol/L | > 250 mg/dL |
| Uric acid | Female: >475.8 μmol/L; | Female: > 8 mg/dL; |
| | Male: >594.8 μmol/L | Male: >10 mg/dL |
| Albumin | <25 g/L | <2.5 g/dL |
| Total bilirubin | $\geq$ 34.2 µmol/L | $\geq$ 2 mg/dL |
| ALT | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| AST | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| Alkaline phosphatase | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| TpI | >ULN | >ULN |
| Methemoglobin | >3.5% | >3.5% |
| BUN | > 17.85 mmol/L | > 50 mg/dL |
| Creatinine | ≥ 177 µmol/L | $\geq$ 2 mg/dL |
| Cholesterol | >10.36 mmol/L | > 400 mg/dL |
| CK | $\geq$ 3 × ULN | $\geq$ 3 × ULN |

| Test | Criteria - System | Criteria – |
|---|---|---|
| | International Units | Conventional Units |
| GGT | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| LDH | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| Phosphorus | < 0.646 mmol/L | Low: <2.0 mg/dL |
| | > 1.777 mmol/L | High: >5.5 mg/dL |
| Urinalysis – Protein | Increase of $\geq 2$ units | Increase of $\geq 2$ units |
| Urinalysis – Glucose | Increase of $\geq 2$ units | Increase of $\geq 2$ units |
| Urinalysis – Blood | Increase of $\geq 2$ units | Increase of $\geq 2$ units |
| Urinalysis – Bilirubin | Increase of $\geq 2$ units | Increase of $\geq 2$ units |

ULN = Upper Limit of Normal

**Appendix C: Criteria for Determining Potentially Clinically Significant Values in Vital Signs** 

| Test | Criteria |
|---|---|
| Systolic Blood Pressure<br>(SBP) – Seated (mmHg) | Increase of $\geq$ 20 mmHg from baseline and $\geq$ 180 mmHg |
| | Decrease of ≥ 20 mmHg from baseline and ≤ 90 mmHg |
| Diastolic Blood Pressure<br>(DBP) – Seated (mmHg) | Increase of $\geq 15$ mmHg from baseline and $\geq 105$ mmHg |
| | <u>Decrease of</u> ≥ 15 mmHg from baseline and ≤50 mmHg |
| Pulse – Seated (beats/min) | Increase of ≥ 15 beats/min from baseline and > 120 beats/min |
| | Decrease of $\geq$ 15 beats/min from baseline and $\leq$ 50 beats/min |
| Temperature | Increase of $\geq 2.0^{\circ}$ C from baseline and $\geq 38.0^{\circ}$ C |
| | Decrease of ≥ 2.0°C from baseline and ≤ 36.0°C |
| Weight | Decrease of $\geq$ 7% from baseline |
| | Decrease of ≥ 10% from baseline |
| | Increase of $\geq$ 7% from baseline |
| | Increase of $\geq 10\%$ from baseline |

# Appendix D: Criteria for Identifying ECG Values that Reflect Potentially Clinically Significant Change

| Parameter | Criterion |
|-------------|----------------------------------------|
| QTcF/QTcB | >470 msec (females), >450 msec (males) |
| PR Interval | >200 msec |
| Heart Rate | <48 |
| | >96 |

## Appendix E: Rules for Determining "Worst" Value

## "Worst" Clinical Laboratory Value

| Rule | Parameters |
|---|---|
| Highest value | Hematology: eosinophils, basophils, monocytes, methemoglobin, reticulocytes |
| | Serum chemistry: ALT, AST, ALK-P, creatinine, total bilirubin, BUN, uric acid, LDH, TSH, creatine kinase, GGT, triglycerides, cholesterol (total) |
| | Urinalysis: all categorical results |
| Lowest value | Hematology: neutrophils, RBC count, HCT, hemoglobin, platelets |
| | Serum chemistry: albumin, creatinine clearance, total protein, oxygen saturation |
| Farthest from | Hematology: WBC count, lymphocytes, MCV, MCH, MCHC |
| normal range<br>midpoint | Serum chemistry: glucose (random), Na, K, phosphate, TBG, T4, calcium, chloride, bicarbonate |
| | Urinalysis: specific gravity, pH |

## "Worst" Vital Sign and Weight Measurement

| Parameter | Criterion for "Worst" Vital Sign |
|--------------------------|-----------------------------------------|
| Systolic blood pressure | Value farthest from 125 mmHg |
| Diastolic blood pressure | Value farthest from 75 mmHg |
| Pulse | Value farthest from 75 beats per minute |
| Respiratory Rate | Highest |
| Weight | Greatest weight loss from baseline |

#### Appendix F: Rules for Scoring the Disease Assessment Scales

#### 1. TPS

Polyp Scoring System Used to Evaluate Polyp Size in Each Nostril by Nasal Endoscopy

| Polyp Score | Polyp Size |
|---|---|
| 0 | No polyps |
| 1 | Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate |
| 2 | Polyps reaching below the lower border of the middle turbinate |
| 3 | Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate |
| 4 | Large polyps causing complete obstruction of the inferior nasal cavity |

Gevaert P, Calus L, Van Zele T, Blomme K, De Ruyck N, Bauters W, et al. Omalizumab is effective in allergic and nonallergic patients with nasal polyps and asthma. J Allergy Clin Immunol 2013;131(1):110-6 e1.

#### 2. The Lund-Mackay scoring system

The Lund-Mackay scoring system as presented in the table below will be used to measure the polyp size in each nostril by computed tomography at all sites except those in the United Kingdom and the Netherlands.

#### **Lund-Mackay Scoring System**

| | Possible Scores <sup>1</sup> |
|---------------------|------------------------------|
| Maxillary | 0-2 |
| Anterior ethmoid | 0-2 |
| Posterior ethmoid | 0-2 |
| Sphenoid | 0-2 |
| Frontal | 0-2 |
| Osteomeatal complex | 0 or 2 |
| Total | |

<sup>1.</sup> Scale: 0 = absence; 1= partial opacification; 2= complete opacification.

#### 3. University of Pennsylvania Smell Identification Test<sup>TM</sup>

The University of Pennsylvania Smell Identification Test consists of 4 booklets, each containing 10 odorants with 1 odorant per page. The stimuli are embedded in plastic microcapsules on brown strips at the bottom of each page. Above each odorant strip is a multiple-choice question with 4 alternative words to describe the odor as in the model of a test page below. The patient is asked to release the odorant by rubbing the brownstrip with the tip of a pencil and to indicate which of 4 words best describes the odor. Thus, each subject receives a score out of 40 possible correct answers (Scadding G, Hellings P, Alobid I, Bachert C, Fokkens W, van Wijk RG, et al. Diagnostic tools in Rhinology EAACI position paper. Clin Transl Allergy 2011;1[1]:2).



Fornazieri MA, Pinna Fde R, Bezerra TF, Antunes MB, Voegels RL. Applicability of the University of Pennsylvania Smell Identification Test (SIT) in Brazilians: pilot study. Braz J Otorhinolaryngol 2010;76(6):695-9.

#### 4. Sino-nasal Outcome Test-22

| I.D.: | SINO-NASAL OUTCOME TEST (SNOT-22) | Date: |
|---|---|---|
| Below you will find a list of symptoms | and social/emotional consequences of your rhinosinusitis. | We would like to know more about |

Below you will find a list of symptoms and social/emotional consequences of your rhinosinusitis. We would like to know more about these problems and would appreciate your answering the following questions to the best of your ability. There are no right or wrong answers, and only you can provide us with this information. Please rate your problems as they have been over the past two weeks. Thank you for your participation. Do not hesitate to ask for assistance if necessary.

| 1. Considering how severe the problem is when you experience it and how often it happens, please rate each item below on how "bad" it is by circling the number that corresponds with how you feel using this scale: → | No Problem | Very Mild Problem | Mild or slight Problem | Moderate Problem | Severe Problem | Problem as bad as it can be | 5 Most Important Items |
|---|---|---|---|---|---|---|---|
| 1. Need to blow nose | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 2. Nasal Blockage | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 3. Sneezing | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 4. Runny nose | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 5. Cough | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 6. Post-nasal discharge | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 7. Thick nasal discharge | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 8. Ear fullness | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 9. Dizziness | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 10. Ear pain | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 11. Facial pain/pressure | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 12. Decreased Sense of Smell/Taste | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 13. Difficulty falling asleep | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 14. Wake up at night | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 15. Lack of a good night's sleep | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 16. Wake up tired | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 17. Fatigue | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 18. Reduced productivity | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 19. Reduced concentration | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 20. Frustrated/restless/irritable | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 21. Sad | 0 | 1 | 2 | 3 | 4 | 5 | 0 |
| 22. Embarrassed | 0 | 1 | 2 | 3 | 4 | 5 | 0 |

<sup>2.</sup> Please mark the most important items affecting your health (maximum of 5 items)

SNOT-20 Copyright © 1996 by Jay F. Piccirillo, M.D., Washington University School of Medicine, St. Louis, Missouri SNOT-22 Developed from modification of SNOT-20 by National Comparative Audit of Surgery for Nasal Polyposis and Rhinosinusitis Royal College of Surgeons of England.

# 5. Visual Analogue Scales for Symptoms of Rhinosinusitis and Clinical Symptoms Improvement Scale

The VASs rank symptoms from 0 (not troublesome) to 10 (most troublesome) on 10 cm-long scales as below.

How troublesome are each of your following symptoms of rhinosinusitus?



Not troublesome Most troublesome









The clinical symptoms improvement scale ranks symptom troublesomeness from 0 (not troublesome) to 10 (worst thinkable troublesome) on a 10 cm-long scale as below.

How troublesome are your symptoms of rhinosinusitis?



The symptomatology or symptom troublesomeness can be divided into "mild," "moderate," and "severe" categories based on total score:

- Mild=0 through 3
- Moderate= >3 through 7
- Severe= >7 through 10

## 6. 36-Item Short Form Health Survey

### SF-36v2 Health Survey Single-Item Presentation Text Standard, United States (English)

Note: Item SF36v2\_BP1 (Item #21) has 6 answers, not 5 answers; see entry for item at end of sheet for more detail.

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 |
|---|---|---|---|---|---|---|---|
| | Your Health and Well-Being | | Score=1 | Score=2 | Score=3 | Score=4 | Score=5 |
| | | This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey! | | | | | |
| | | For each of the following questions, please select the one box that best describes your answer. | | | | | |
| SF36v2_GH1 | None | In general, would you say your health is: | Excellent | Very good | Good | Fair | Poor |
| SF36v2_HT | None | Compared to one year ago, how would you rate your health in general now? | Much<br>better<br>now than<br>one year<br>ago | Somewhat<br>better now<br>than one<br>year ago | About the same as one year ago | Somewhat<br>worse<br>now than<br>one year<br>ago | Much<br>worse<br>now than<br>one year<br>ago |
| SF36v2_PF01 | The following question is about activities you might do during a typical day. | Does your health now limit you in vigorous activities, such as running, lifting heavy objects, participating in strenuous sports? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all | | |
| SF36v2_PF02 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in <u>moderate</u> <u>activities</u> , such as moving a table, pushing a vacuum cleaner, bowling, or playing golf? If | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all | | |

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 |
|---|---|---|---|---|---|---|---|
| | | so, how much? | | | | | |
| SF36v2_PF03 | The following question is about activities you might do during a typical day. | Does your health now limit you in lifting or carrying groceries? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all | | |
| SF36v2_PF04 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in climbing <u>several</u> flights of stairs? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all | | |
| SF36v2_PF05 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in climbing <u>one</u> flight of stairs? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not limited at all | | |
| SF36v2_PF06 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in bending, kneeling, or stooping? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not limited at all | | |
| SF36v2_PF07 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in walking <u>more</u> <u>than a mile</u> ? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not limited at all | | |
| SF36v2_PF08 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in walking <u>several hundred yards</u> ? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all | | |
| SF36v2_PF09 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in walking <u>one</u> <u>hundred yards</u> ? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all | | |
| SF36v2_PF10 | The following question is about activities you might do during a typical day. | Does <u>your health now limit you</u> in bathing or dressing yourself? If so, how much? | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not limited at all | | |
| SF36v2_RP1 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Cut down on the <u>amount of time</u> you spent on work or other activities <u>as a result of your physical health</u> | All of the time | Most of the time | Some of the time | A little of the time | None of the time |

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 |
|---|---|---|---|---|---|---|---|
| SF36v2_RP2 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Accomplished less than you would like as a result of your physical health | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_RP3 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Were limited in the kind of work or other activities as a result of your physical health | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_RP4 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Had <u>difficulty</u> performing the work or other activities <u>as a result of your physical health</u> (for example, it took extra effort) | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_RE1 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Cut down on the <u>amount of time</u> you spent on work or other activities <u>as a result of any</u> <u>emotional problems</u> (such as feeling depressed or anxious) | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_RE2 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Accomplished less than you would like as a result of any emotional problems (such as feeling depressed or anxious) | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_RE3 | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities? | Did work or other activities <u>less carefully than</u> <u>usual as a result of any emotional problems</u> (such as feeling depressed or anxious) | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_SF1 | None | During the <u>past 4 weeks</u> , to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? | Not at all | Slightly | Moderately | Quite a bit | Extremely |
| SF36v2_BP1 | None | How much <u>bodily</u> pain have you had during the <u>past 4 weeks?</u> | | See end of o | l<br>document for a | nswers #1-#6 | 1 |

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 |
|---|---|---|---|---|---|---|---|
| SF36v2_BP2 | None | During the <u>past 4 weeks</u> , how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)? | Not at all | A little bit | Moderately | Quite a bit | Extremely |
| SF36v2_VT1 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks did you feel full of life? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_MH1 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks have you been very nervous? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_MH2 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the <u>past 4 weeks</u> have you felt so down in the dumps that nothing could cheer you up? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_MH3 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks have you felt calm and peaceful? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_VT2 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks did you have a lot of energy? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_MH4 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been | How much of the time during the <u>past 4 weeks</u> have you felt downhearted and depressed? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 |
|---|---|---|---|---|---|---|---|
| | feeling. | | | | | | |
| SF36v2_VT3 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks did you feel worn out? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_MH5 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks have you been happy? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_VT4 | This question is about how you feel and how things have been with you during the past 4 weeks. Please give the one answer that comes closest to the way you have been feeling. | How much of the time during the past 4 weeks did you feel tired? | All of the time | Most of<br>the time | Some of the time | A little of the time | None of the time |
| SF36v2_SF2 | None | During the <u>past 4 weeks</u> , how much of the time has your <u>physical health or emotional</u> <u>problems</u> interfered with your social activities (like visiting with friends, relatives, etc.)? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| SF36v2_GH2 | How TRUE or FALSE is the following statement for you? | I seem to get sick a little easier than other people. | Definitely<br>true | Mostly<br>true | Don't know | Mostly<br>false | Definitely false |
| SF36v2_GH3 | How TRUE or FALSE is the following statement for you? | I am as healthy as anybody I know. | Definitely<br>true | Mostly<br>true | Don't know | Mostly false | Definitely false |
| SF36v2_GH4 | How TRUE or FALSE is the following statement for you? | I expect my health to get worse. | Definitely<br>true | Mostly<br>true | Don't know | Mostly<br>false | Definitely false |
| SF36v2_GH5 | How TRUE or FALSE is the following statement for you? | My health is excellent. | Definitely true | Mostly<br>true | Don't know | Mostly false | Definitely false |

#### Data for item SF36v2\_BP1 (item #21 in the survey template)

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 | Answer<br>Text 6 |
|---|---|---|---|---|---|---|---|---|
| SF36v2_BP1 | None | How much <u>bodily</u> pain have you had during the<br><u>past 4 weeks</u> ? | None | Very mild | Mild | Moderate | Severe | Very severe |

SF-36v2® Health Survey Ó 1992, 1996, 2000, 2010 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved.

(SF-36v2® Health Survey Single-Item Presentation Text Standard, United States (English))

SF-36® is a registered trademark of Medical Outcomes Trust.

## 7. Asthma Control Test<sup>TM</sup>

# Asthma Control Test™ Single-Item Presentation Text, United States (English)

| Item Name | Instructions | Question Text | Answer<br>Text 1 | Answer<br>Text 2 | Answer<br>Text 3 | Answer<br>Text 4 | Answer<br>Text 5 |
|---|---|---|---|---|---|---|---|
| | Asthma Control Test™ | | | | | | |
| | This survey was designed to help you describe your asthma and how your asthma affects how you feel and what you are able to do. For each of the following questions, please select the one box that best describes your answer. | | | | | | |
| ACT1 | None | In the <u>past 4 weeks</u> , how much of the time did your <u>asthma</u> keep you from getting as much done at work, school or at home? | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| ACT2 | None | During the <u>past 4 weeks</u> , how often have you had shortness of breath? | More than once a day | Once a<br>day | 3 to 6<br>times a<br>week | Once or<br>twice<br>a week | Not at all |
| ACT3 | None | During the <u>past 4 weeks</u> , how often did your <u>asthma</u> symptoms (wheezing, coughing, shortness of breath, chest tightness or pain) wake you up at night or earlier than usual in the morning? | 4 or more<br>nights a<br>week | 2 to 3<br>nights a<br>week | Once a<br>week | Once or<br>Twice | Not at all |
| ACT4 | None | During the <u>past 4 weeks</u> , how often have you used your rescue inhaler or nebulizer medication (such as Albuterol, Ventolin®, Proventil®, or Maxair®)? | 3 or more<br>times per<br>day | 1 or 2<br>times per<br>day | 2 or 3<br>times per<br>week | Once a<br>week<br>or less | Not at all |
| ACT5 | None | How would you rate your <u>asthma</u> control during the <u>past 4 weeks?</u> | Not<br>Controlled<br>at all | Poorly<br>Controlled | Somewhat<br>Controlled | Well<br>Controlled | Completely Controlled |

Asthma Control Test<sup>TM</sup> © QualityMetric Incorporated 2002, 2004, 2011. All rights reserved. Asthma Control Test<sup>TM</sup> is a trademark of QualityMetric Incorporated.

Single-Item Presentation Text, United States (English)

## Appendix G: List of Review Files Provided by Allakos to InClin

- 1. Protocol deviations identified by subject and a flag per each deviation type.
- 2. Coding or coding advice on any concomitant medication or adverse event that requires special review and input from Allakos or per the DMC.

## Appendix H: List of Tables, Figures, and Listings

## **List of Tables**

| Table | |
|---|---|
| Number | Table Description |
| 14.1.1.1 | Subject Disposition (All Subjects) |
| 14.1.1.2 | Subject Disposition by Region (All Subjects) |
| 14.1.2.1 | Early Discontinuation of Study Drug by Time Period (Safety Population) |
| 14.1.2.2 | Early Discontinuation of Study Drug by Time Period (MITT Population) |
| 14.1.3 | Protocol Deviations (MITT Population) |
| 14.1.4.1 | Demographic and Baseline Characteristics (Safety Population) |
| 14.1.4.2 | Demographic and Baseline Characteristics (MITT Population) |
| 14.1.4.3 | Demographic and Baseline Characteristics by Region (MITT Population) |
| 14.1.5 | Medical History at Baseline (Safety Population) |
| 14.1.6 | Baseline Physical and Neurological Examination (Safety Population) |
| 14.1.7.1 | Prior Medications (Safety Population) |
| 14.1.7.2.1 | Concomitant Medications (Safety Population) |
| 14.1.7.2.2 | Concomitant Medications (MITT Population) |
| 14.1.7.3 | Study Drug Administration (Safety Population) |
| 14.2.8.1 | Change in Total Polyp Score (TPS) from Baseline to Week 12 (No |
| | Imputation) (MITT Population) |
| 14.2.8.2 | Change in Total Polyp Score (TPS) from Baseline to Week 12 (With |
| | Imputation ) (MITT Population) |
| 14.2.8.3 | Change in Total Polyp Score (TPS) from Baseline to Week 12 (No |
| | Imputation) (ITT Population) |
| 14.2.8.4 | Change in Total Polyp Score (TPS) from Baseline to Week 12 (No |
| | Imputation) (PP Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.2.9.1 | Change in Total Polyp Score (TPS) from Baseline over Time (No |
| | Imputation) (MITT Population) |
| 14.2.9.2 | Change in Total Polyp Score (TPS) from Baseline over Time (With |
| | Imputation) (MITT Population) |
| 14.2.9.3 | Change in Total Polyp Score (TPS) from Baseline over Time (No |
| | Imputation) (ITT Population) |
| 14.2.9.4 | Change in Total Polyp Score (TPS) from Baseline over Time (No |
| | Imputation) (PP Population) |
| 14.2.9.5 | Change in Total Polyp Score (TPS) from Baseline over Time (Without |
| | Time Interaction) (MITT Population) |
| 14.2.9.6 | Percent Change in Total Polyp Score (TPS) from Baseline over Time |
| | (Without Time Interaction) (MITT Population) |
| 14.2.9.7 | Absolute Measurements in Total Polyp Score (TPS) from Baseline over |
| | Time (Without Time Interaction) (MITT Population) |
| 14.2.9.8 | Total Polyp Score (TPS) – Time to Response at Any Time (MITT |
| | Population) |
| 14.2.10.1 | Subgroup Analysis of TPS Score at Week 12 by Gender (MITT |
| | Population) |
| 14.2.10.2 | Subgroup Analysis of TPS Score at Week 12 by Age (MITT Population) |
| 14.2.10.3 | Subgroup Analysis of TPS Score at Week 12 by Asthma (MITT |
| | Population) |
| 14.2.10.4 | Subgroup Analysis of TPS Score at Week 12 by 1-point Reduction |
| | Responder Criteria (MITT Population) |
| 14.2.10.5 | Subgroup Analysis of TPS Score at Week 12 by 20% Reduction |
| | Responder Criteria (MITT Population) |
| 14.2.10.6 | Subgroup Analysis of TPS Score at Week 12 by 30% Reduction |
| | Responder Criteria (MITT Population) |
| 14.2.11 | Change in Size of Polyps (Lund-Mackay Score) from Baseline to Week |
| | 12 (MITT Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.2.12.1 | Change in Peak Nasal Inspiration Flow (PNIF) from Baseline over Time |
| | (MITT Population) |
| 14.2.12.2 | Peak Nasal Inspirational Flow (PNIF) – Time to Response at Any Time |
| | (MITT Population) |
| 14.2.13.1 | Change in Sense of Smell (UPSIT Total Score) from Baseline over Time (MITT Population) |
| 14.2.13.2 | Sense of Smell (UPSIT) – Time to Response at Any Time (MITT |
| | Population) |
| 14.2.14.1 | Sino-nasal Outcome Test-22 (SNOT-22) (Five Most Important Items) at Week 12 (MITT Population) |
| 14.2.14.2 | Change in SNOT-22 (Total Score of Five Most Important Items) from |
| | Baseline over Time (MITT Population) |
| 14.2.14.3 | Change in SNOT-22 (Total Score of All Items) from Baseline over Time |
| | (MITT Population) |
| 14.2.14.4 | Sino-nasal Outcome Test-22 (SNOT-22) – Time to Response at Any |
| | Time (MITT Population) |
| 14.2.15.1 | Visual Analogue Scale (VAS) by Symptom (MITT Population) |
| 14.2.15.2 | Change in Visual Analogue Scale (VAS by Symptom) from Baseline over Time (MITT Population) |
| 14.2.15.3 | Change in Visual Analogue Scale (VAS Total Score) from Baseline over Time (MITT Population) |
| 14.2.15.4 | Visual Analogue Scale (VAS) – Time to Response at Any Time (MITT Population) |
| 14.2.15.5 | Change in Clinical Symptoms Improvement Scale (Total Score) from |
| | Baseline over Time (MITT Population) |
| 14.2.16 | Change in 36-Item Short Form Health Survey (SF-36 Total Score) from |
| | Baseline over Time (MITT Population) |
| 14.2.17.1 | Biomarker Analysis: Change in Biomarkers from Baseline Over Time |
| | (Biomarker Population, Sub-Study) |

| Table | |
|---|---|
| Number | Table Description |
| 14.2.17.2 | Biomarker Analysis: Percent Change in Biomarkers from Baseline over |
| | Time (Biomarker Population, Sub-Study) |
| 14.2.17.3 | Biomarker Analysis: Change in Biomarkers from Baseline over Time |
| | (Biomarker Population, All Patients) |
| 14.2.17.4 | Biomarker Analysis: Percent Change in Biomarkers from Baseline over |
| | Time (Biomarker Population, All Patients) |
| 14.2.18.1 | Change in Forced Expiratory Volume in 1 Second (FEV1) from Baseline |
| | to Week 7 (MITT Population in Patients with Comorbid Asthma) |
| 14.2.18.2 | Change in Forced Vital Capacity (FVC) from Baseline to Week 7 (MITT |
| | Population in Patients with Comorbid Asthma) |
| 14.2.18.3 | Change in Forced Expiratory Flow (FEF) from Baseline to Week 7 |
| | (MITT Population in Patients with Comorbid Asthma) |
| 14.2.18.4 | Change in Asthma Control Test (ACT) from Baseline to Week 12 (MITT |
| | Population in Patients with Comorbid Asthma) |
| 14.2.18.5.1 | Use of Asthma Rescue Therapy from Baseline to Week 12 (MITT |
| | Population in Patients with Comorbid Asthma) |
| 14.2.18.5.2 | Use of Asthma Rescue Therapy - Shift from Baseline to Week 12 (MITT |
| | Population in Patients with Comorbid Asthma) |
| 14.3.1.19.1 | Overall Summary of All Adverse Events (Safety Population) |
| 14.3.1.19.2. | Treatment-Emergent Adverse Events by System Organ Class and |
| 1 | Preferred Term (Safety Population) |
| 14.3.1.19.2. | Treatment-Emergent Adverse Events by System Organ Class, Preferred |
| 2 | Term and Severity (Safety Population) |
| 14.3.1.19.2. | Treatment-Emergent Adverse Events by System Organ Class, Preferred |
| 3 | Term and Relationship to Study Drug (Safety Population) |
| 14.3.2.19.3 | Treatment-Emergent Serious Adverse Events by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.19.4. | Treatment-Emergent Fatal Serious Adverse Events by System Organ |
| 1 | Class and Preferred Term (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.19.4. | Treatment-Emergent Non-Fatal Serious Adverse Events by System Organ |
| 2 | Class and Preferred Term (Safety Population) |
| 14.3.1.19.5 | Treatment-Emergent Severe Adverse Events by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.1.19.6 | Day 0 Treatment Emergent Adverse Events by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.1.19.7 | Post-Treatment Adverse Events by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.1.19.8. | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety |
| 1 | Population Subgroup: Asthma Present) |
| 14.3.1.19.8. | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety |
| 2 | Population Subgroup: Asthma Absent) |
| 14.3.1.19.8. | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety |
| 3 | Population Subgroup: Using Concomitant Medication at Any Time |
| | During the Study) |
| 14.3.1.19.8. | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety |
| 4 | Population Subgroup: Not Using Concomitant Medication at Any Time |
| | During the Study) |
| 14.3.1.19.8. | Treatment-Emergent Adverse Events by SOC and Preferred Term in at |
| 5 | least 5 Subjects in any of Treatment Group (Safety Population) |
| 14.3.4.20.1. | Hematology Values and Changes from Baseline at All Visits – |
| 1 | Conventional Units (Safety Population) |
| 14.3.4.20.1. | Hematology Values and Changes from Baseline at All Visits – SI Units |
| 2 | (Safety Population) |
| 14.3.4.20.1. | Hematology – Shift from Baseline (Safety Population) |
| 3 | |
| 14.3.4.20.2. | Serum Chemistry Values and Changes from Baseline at All Visits – |
| 1 | Conventional Units (Safety Population) |
| 14.3.4.20.2. | Serum Chemistry Values and Changes from Baseline at All Visits – SI |
| 2 | Units (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.4.20.2. | Serum Chemistry – Shift from Baseline (Safety Population) |
| 3 | |
| 14.3.4.20.3. | Urinalysis Values at All Visits – (Safety Population) |
| 1 | |
| 14.3.4.20.3. | Urinalysis – Shift from Baseline (Part 1 of 2) (Safety Population) |
| 2.1 | |
| 14.3.4.20.3. | Urinalysis – Shift from Baseline (Part 2 of 2) (Safety Population) |
| 2.2 | |
| 14.3.4.21.1 | Vital Signs – Day 0 Pre-Dose and Post-Dose (Safety Population) |
| 14.3.4.21.2 | Vital Signs – Screening and Post Day 0 (Safety Population) |
| 14.3.4.21.3 | Incidence of Potentially Clinically Significant Vital Sign Results (Safety |
| | Population) |

# **List of Figures**

| Figure | |
|---|---|
| Number | Figure Description |
| 14.2.1.1 | Least Squares Mean Change in Total Polyp Score (TPS) (MITT |
| | Population) |
| 14.2.1.2 | Least Squares Mean Change in Total Polyp Score (TPS) (MITT |
| | Population in Patients with Comorbid Asthma) |
| 14.2.1.3 | Kaplan-Meier Curves for Time to 1-point Reduction in Total Polyp Score |
| | (TPS) (MITT Population) |
| 14.2.2 | Least Squares Mean Change in Peak Nasal Inspiratory Flow (PNIF) |
| | (MITT Population) |
| 14.2.3 | Least Squares Mean Change in University of Pennsylvania Smell |
| | Identification Test (UPSIT) (MITT Population) |
| 14.2.4 | Least Squares Mean Change in 22-item Sinonasal Outcome Test (SNOT- |
| | 22) (MITT Population) |
| 14.2.5 | Least Squares Mean Change in Visual Analogue Scale (VAS) (MITT |
| | Population) |
| 14.2.6 | Least Squares Mean Change in Forced Expiratory Volume in 1 Second |
| | (FEV1) (MITT Population in Patients with Comorbid Asthma) |
| 14.2.7 | Least Squares Mean Change in Asthma Control Test (ACT) (MITT |
| | Population in Patients with Comorbid Asthma) |
| 14.2.8 | Least Squares Mean Change in Blood Eosinophil Count (Biomarker |
| | Population) |

# **List of Data Listings**

| Listing | |
|---|---|
| Number | Listing Description |
| 16.2.1.1.1 | Subject Populations |
| 16.2.1.1.2 | Subject Disposition |
| 16.2.1.1.3 | Subject Visit Dates |
| 16.2.2.2 | Protocol Deviations |
| 16.2.2.3 | Inclusion/Exclusion Findings |
| 16.2.1.4.1 | Informed Consent |
| 16.2.1.4.2 | Withdrawal of Consent |
| 16.2.4.5.1 | Demographics and Baseline Characteristics (Part 1 of 2) |
| 16.2.4.5.2 | Demographics and Baseline Characteristics (Part 2 of 2) |
| 16.2.4.6 | Relevant Respiratory History at Screening |
| 16.2.4.7 | Medical History at Screening |
| 16.2.4.8 | Physical and Neurological Examination |
| 16.2.4.9 | Symptom Directed Physical Examination |
| 16.2.4.10 | Electrocardiogram at Screening |
| 16.2.4.11.1 | Pregnancy Test |
| 16.2.4.11.2 | Pregnancy Report during Study |
| 16.2.4.12 | Follicle-Stimulating Hormone (FSH) Test at Screening |
| 16.2.4.13 | Fecal Sample Test at Screening |
| 16.2.4.14 | Anti-Drug Antibody (ADA) |
| 16.2.4.15 | Exploratory Biomarkers |
| 16.2.4.16 | Serum Samples for Total Immunoglobulin E and ImmunoCAP on Day -3 |
| 16.2.4.17 | Prior Medications |
| 16.2.4.18 | Concomitant Medications |
| 16.2.4.19 | Intranasal Steroid Adjustment at Day 0 |
| 16.2.5.20 | Study Drug Administration |

| Listing | |
|---|---|
| Number | Listing Description |
| 16.2.6.21.1 | Total Polyp Score (TPS) |
| 16.2.6.21.2 | Size of Polyps (Lund-Mackay Score) |
| 16.2.6.21.3 | Peak Nasal Inspiratory Flow (PNIF) |
| 16.2.6.21.4 | University of Pennsylvania Smell Identification Test (UPSIT) |
| 16.2.6.21.5 | Sino-nasal Outcome Test-22 (SNOT-22) |
| 16.2.6.21.6 | Visual Analogue Scale (VAS) |
| 16.2.6.21.7 | Clinical Symptoms Improvement Scale |
| 16.2.6.21.8.1 | 36-Item Short Form Health Survey (SF-36) (Part 1 of 3) |
| 16.2.6.21.8.2 | 36-Item Short Form Health Survey (SF-36) (Part 2 of 3) |
| 16.2.6.21.8.3 | 36-Item Short Form Health Survey (SF-36) (Part 3 of 3) |
| 16.2.6.21.9 | Asthma Control Test (ACT) |
| 16.2.6.21.10 | Spirometry Test |
| 16.2.6.21.11.1 | Sub-study Biomarkers (Part 1 of 2) |
| 16.2.6.21.11.2 | Sub-study Biomarkers (Part 2 of 2) |
| 16.2.7.22.1 | Adverse Events |
| 16.2.7.22.2 | Treatment-Emergent Serious Adverse Events (Collected on AE CRF) |
| 16.2.7.22.3 | Fatal Treatment-Emergent Serious Adverse Events (Collected on AE |
| | CRF) |
| 16.2.7.22.4 | Non-Fatal Treatment-Emergent Serious Adverse Events (Collected on AE |
| | CRF) |
| 16.2.8.23.1.1 | Central Laboratory Normal Ranges – Conventional Units |
| 16.2.8.23.1.2 | Central Laboratory Normal Ranges – SI Units |
| 16.2.8.23.2.1 | Hematology – Conventional Units (Part 1 of 2) |
| 16.2.8.23.2.2 | Hematology – Conventional Units (Part 2 of 2) |
| 16.2.8.23.2.3 | Hematology – SI Units |
| 16.2.8.23.3.1 | Serum Chemistry – Conventional Units (Part 1 of 2) |
| 16.2.8.23.3.2 | Serum Chemistry – Conventional Units (Part 2 of 2) |
| 16.2.8.23.3.3 | Serum Chemistry – SI Units |
| 16.2.8.23.4 | Urinalysis |

| Listing<br>Number | Listing Description |
|-------------------|-------------------------------------------------------|
| 16.2.8.24.1 | Vital Signs |
| 16.2.8.24.2 | Vital Sign Results of Potential Clinical Significance |

**Appendix I: Table Layouts** 

**Table 14.1.1.1 Subject Disposition** All Subjects

| | DI I | AK001 | AK001 | AK001 | T . 1 |
|---|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined | Total |
| Subjects Screened | | | | | n |
| Subjects Randomized [1] | n | n | n | n | n |
| Safety Population [2] | n (%) | n (%) | n (%) | n (%) | n (%) |
| ITT Population [3] | n (%) | n (%) | n (%) | n (%) | n (%) |
| MITT Population [4] | n (%) | n (%) | n (%) | n (%) | n (%) |
| PP Population [5] | n (%) | n (%) | n (%) | n (%) | n (%) |
| Completed Study | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| Completed study and completed treatment | n (%) | n (%) | n (%) | n (%) | n (%) |
| Completed study but off treatment | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| All Reasons for Study Drug Discontinuation | | | | | |
| Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| All Reasons for Study Discontinuation [6] | | | | | |
| Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Primary Reason for Study Discontinuation | | | | | |
| Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | . , | . , | • • | ` ′ | . , |


<sup>[1]</sup> All percentages are based on the number of subjects randomized. [2] All randomized subjects who take at least one dose of study drug.

<sup>[3]</sup>All randomized subjects.

<sup>[4]</sup> All randomized subjects who take at least one dose of the study drug and have both a baseline and at least one post-baseline effifcay assessment. [5] All MITT population subjects who have a week 12 visit and valid efficacy measurements. [6] Subjects may be counted for more than one reason for study discontinuation but are counted only once for primary reason for discontinuation.

| Note: The following 5 subjects vvv, www, xxx, yyy, zzz were randomized but n | ot dosed. (programming note: List the subject IDs | <i>s</i> ) |
|---|---|---|
| ak001-002_statistical analysis plan_final_v1_2017_08_16 | | CONFIDENTIAL |

Table 14.1.1.2 Subject Disposition by Region All Subjects

| Danian | | Dlasaka | AK001 | AK001 | AK001 | T-4-1 |
|---|---|---|---|---|---|---|
| Region | | Placebo | 25 mg | 250 mg | Combined | Total |
| United States | Subjects Screened | | | | | n |
| | Subjects Randomized [1] | n | n | n | n | n |
| | Safety Population [2] | n (%) | n (%) | n (%) | n (%) | n (%) |
| | ITT Population [3] | n (%) | n (%) | n (%) | n (%) | n (%) |
| | MITT Population [4] | n (%) | n (%) | n (%) | n (%) | n (%) |
| | PP Population [5] | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Completed Study | | | | | |
| | Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Completed study and completed treatment | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Completed study but off treatment | n (%) | n (%) | n (%) | n (%) | n (%) |
| | No | n (%) | n (%) | n (%) | n (%) | n (%) |
| | All Reasons for Study Drug Discontinuation | | | | | |
| | Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | All Reason for Study Discontinuation [6] | | | | | |
| | Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Primary Reason for Study Discontinuation | | | | | |
| | Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | ` / | . , | ` / | , | ` ' |

European Union

. . .
Note: The following 5 subjects vvv, www, xxx, yyy, zzz were randomized but not dosed. (programming note: List the subject IDs)

path\t program.sas date time

Programming note: Start each region on a new page.

<sup>[1]</sup> Percentages for screen failures are based on the number of subjects screened – subjects may be counted in multiple screen failure categories. All other percentages are based on the number of subjects randomized.

<sup>[2]</sup> All randomized subjects who take at least one dose of study drug.

<sup>[3]</sup> All randomized subjects.

<sup>[4]</sup> All randomized subjects who take at least one dose of the study drug and have both a baseline and at least one post-baseline effifcay assessment.

<sup>[5]</sup> All MITT population subjects who have a week 12 visit and valid efficacy measurements.

<sup>[6]</sup> Subjects may be counted for more than one reason for study discontinuation but are counted only once for primary reason for discontinuation.

Table 14.1.2.1
Early Discontinuation of Study Drug by Time Period
Safety Population

| Subjects Taking at Least One Dose Early Discontinuation of Study Drug [1] Early Discontinuation of Study Drug before Day 14 | Placebo n n (%) | 25 mg n n (%) | 250 mg<br>n<br>n (%) | n n (%) | Total<br>n<br>n (%) |
|---|---|---|---|---|---|
| Early Discontinuation of Study Drug [1] Early Discontinuation of Study Drug before Day 14 | n (%) | n (%) | | | |
| Early Discontinuation of Study Drug before Day 14 | | | n (%) | n (%) | n (%) |
| Day 14 | n (%) | n (%) | | | |
| | | n (%) | n (%) | n (%) | n (%) |
| Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| ••• | | | | | |
| Early Discontinuation of Study Drug During<br>Days >14-21 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| ••• | | | | | |
| Early Discontinuation of Study Drug During Days >21-49 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) | n (%) | n (%) |

Note: Percentages are based on the number of subjects in the Safety Population.

[1] Drug discontinuation prior to Week 12 will be considered early.

path\t\_program.sas date time

Programming note: Repeat this table for MITT population (Table 14.1.2.2)

Table 14.1.3 Protocol Deviations MITT Population

| | Placebo | AK001<br>25 mg | AK001<br>250 mg | AK001<br>Combined | Total |
|---|---|---|---|---|---|
| | (N=) | (N= ) | (N=) | (N=) | (N= ) |
| All Deviations | n (%) | n (%) | n (%) | n (%) | n (%) |
| Informed consent | n (%) | n (%) | n (%) | n (%) | n (%) |
| Randomization error | n (%) | n (%) | n (%) | n (%) | n (%) |
| Safety | n (%) | n (%) | n (%) | n (%) | n (%) |
| Efficacy | n (%) | n (%) | n (%) | n (%) | n (%) |
| IP/Treatment deviation | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other deviations | n (%) | n (%) | n (%) | n (%) | n (%) |
| Type of Protocol Deviation [1] | | | | | |
| Informed consent procedures | n (%) | n (%) | n (%) | n (%) | n (%) |
| Eligibility criteria | n (%) | n (%) | n (%) | n (%) | n (%) |
| Study procedure not done | n (%) | n (%) | n (%) | n (%) | n (%) |
| Study procedure not per protocol | n (%) | n (%) | n (%) | n (%) | n (%) |
| Patient not withdrawn as per protocol | n (%) | n (%) | n (%) | n (%) | n (%) |
| Study drug administration | n (%) | n (%) | n (%) | n (%) | n (%) |
| Missed study visit | n (%) | n (%) | n (%) | n (%) | n (%) |
| Visit out of study window | n (%) | n (%) | n (%) | n (%) | n (%) |
| Safety reporting | n (%) | n (%) | n (%) | n (%) | n (%) |
| Prohibited con meds/therapies | n (%) | n (%) | n (%) | n (%) | n (%) |
| Laboratory samples | n (%) | n (%) | n (%) | n (%) | n (%) |
| Study drug storage and handling | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other deviations | n (%) | n (%) | n (%) | n (%) | n (%) |

[1] All categories include that fall under the "other" category

path\t\_program.sas date time

Programming note: The categories in first column should come from SAP section 7.2

Table 14.1.4.1
Demographic and Baseline Characteristics
Safety Population

| | | AK001 | AK001 | AK001 | |
|---|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined | Total |
| | (N=) | (N= ) | (N=) | (N=) | (N= ) |
| Age at Informed Consent (years) | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | xx, xx |
| < Median | n (%) | n (%) | n (%) | n (%) | n (%) |
| $\geq$ Median | n (%) | n (%) | n (%) | n (%) | n (%) |
| Gender | | | | | |
| Male | n (%) | n (%) | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ethnicity | | | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) |
| Race | | | | | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) | n (%) | n (%) |
| Black or African American | n (%) | n (%) | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) |
| Geographic Region | | | | | |
| United States | n (%) | n (%) | n (%) | n (%) | n (%) |
| European Union | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t\_program.sas date time *Table continues on next page*.

Table 14.1.4.1 Demographic and Baseline Characteristics Safety Population (cont'd)

| | | AK001 | AK001 | AK001 | |
|---|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined | Total |
| | (N=) | (N= ) | (N=) | (N=) | (N= ) |
| Subject Consented | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Height (cm) | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx, xx |
| Weight (kg) | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx, xx |
| BMI (kg/m <sup>2</sup> ) | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX, XX |

path\t\_program.sas date time

Programming note: Repeat table for MITT Population (Table 14.1.4.2).

**Table 14.1.4.3** Demographic and Baseline Characteristics by Region **MITT Population** 

| Region | | Placebo<br>(N=) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) | Total<br>(N= ) |
|---|---|---|---|---|---|---|
| United States | Age at Informed Consent (years) | | | | | |
| Office States | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X (XX.XX) | XX.X (XX.XX) | XX.X | XX.X | XX.X (XX.XX) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | < Median | n (%) | n (%) | n (%) | n (%) | n (%) |
| | ≥ Median | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Gender | | | | | |
| | Male | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Female | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Ethnicity | | | | | |
| | Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Not Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) |
| | ••• | | | | | |
| European Union | | | | | | |

path\t\_program.sas date time

Programming note: See previous mock table for variables to include. Exclude Geographic Region.

Table 14.1.5 Medical History at Baseline Safety Population

| | | AK001 | AK001 | AK001 | |
|---|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined | Total |
| MedDRA System Organ Class | (N=) | (N=) | (N=) | (N=) | (N= ) |
| Blood and Lymphatic System Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cardiac Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Congenital, Familial and Genetic Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ear and Labyrinth Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Endocrine Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Eye Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Gastrointestinal Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| General Disorders and Administration Site | n (%) | n (%) | n (%) | n (%) | n (%) |
| Conditions | | | | | |
| Hepatobiliary Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| mmune System Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| Infections and Infestations | n (%) | n (%) | n (%) | n (%) | n (%) |
| njury, Poisoning and Procedural | n (%) | n (%) | n (%) | n (%) | n (%) |
| Complications | , | ` / | . , | . , | , , |
| nvestigations | n (%) | n (%) | n (%) | n (%) | n (%) |
| Metabolism and Nutrition Disorders | n (%) | n (%) | n (%) | n (%) | n (%) |
| etc. | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Programming note: Sort table based on SOC order alphabetically

Table 14.1.6

Baseline Physical and Neurological Examination
Safety Population

| Body System | Findings | Placebo<br>(N= ) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) | Total<br>(N= ) |
|---|---|---|---|---|---|---|
| Skin | | | | | | |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Abnormal NCS | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Abnormal CS | n (%) | n (%) | n (%) | n (%) | n (%) |
| Head | | | | | | |

Note: NCS = Not clinically significant, CS = Clinically significant.

path\t program.sas date time

Programming note: Table will include all physical examination body systems in SAP section 7.5: Skin, Head, Eyes, Ears, Nose, Throat, Thyroid, Lungs, Cardiovascular system, Abdomen, Extremities, Lymph nodes and neurological examination.

**Table 14.1.7.1 Prior Medications Safety Population** 

| D1 1 | | AK001 | AK001 | |
|---|---|---|---|---|
| Placebo | 25 mg | 250 mg | Combined | Total |
| (N=) | (N= ) | (N=) | (N=) | (N= ) |
| n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) | n (%) | n (%) n (%) n (%) n (%) n (%) n (%) n (%) n (%) |

Prior medications are those that started within the 30 days before Screening.

Note: At each level of summation (overall, ATC classes, generic drug name), subjetcs reporting more than once of the same medication are counted only once for a particular medication class and medication. Each summary is ordered alphabetically by ATC class and generic drug name within each ATC class.

path\t program.sas date time

Table 14.1.7.2.1 Concomitant Medications Safety Population

| ATC Class (Level 1) / | | AK001 | AK001 | AK001 | |
|---|---|---|---|---|---|
| ATC Class (Level 3)/ | Placebo | 25 mg | 250 mg | Combined | Total |
| Generic Drug Name | (N=) | (N= ) | (N=) | (N=) | (N= ) |
| Subjects Receiving Concomitant <sup>[1]</sup> Medications | n (%) | n (%) | n (%) | n (%) | n (%) |
| ATC Class (Level 1) 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| ATC Class (Level 3) 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Generic Drug Name 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Generic Drug Name 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| ATC Class (Level 3) 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Generic Drug Name 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Generic Drug Name 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| ATC Class (Level 1) 2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| ATC Class (Level 3) 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Generic Drug Name 1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Generic Drug Name 2 | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Concomitant medications are those medications taken at the start of study drug or initiated after the initial dose of study drug.

Note: At each level of summation (overall, ATC classes, generic drug name), subjects reporting more than once of the same medication are counted only once for a particular medication class and medication. Each summary is ordered alphabetically by ATC class and generic drug name within each ATC class.

path\t program.sas date time

Programming note: Repeat table for MITT Population (Table 14.1.7.2.2). Programming note: Separate prior meds and concomitant meds (2 tables)

Table 14.1.7.3 Study Drug Administration Safety Population

| | | Placebo | AK001<br>25 mg | AK001<br>250 mg | AK001<br>Combined |
|---|---|---|---|---|---|
| Time Point | | (N=) | (N= ) | (N=) | (N=) |
| Day 0 | Arm for Infusion | (0/) | (0/) | (0/) | (0/) |
| | Left Arm | n (%) | n (%) | n (%) | n (%) |
| | Right Arm | n (%) | n (%) | n (%) | n (%) |
| | Full Infusion Given | | | | |
| | Yes | n (%) | n (%) | n (%) | n (%) |
| | No | n (%) | n (%) | n (%) | n (%) |
| | If Yes, Total Volume of Study Drug<br>Administered (mL) | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX | XX, XX |
| | If No, Total Amount Given (mL) | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX | xx, xx |
| | Infusion Interrupted | | | | |
| | Yes | n (%) | n (%) | n (%) | n (%) |
| | No | n (%) | n (%) | n (%) | n (%) |
| | If Yes, Number of Times Interrupted | , | | . , | , |
| | 1 | n (%) | n (%) | n (%) | n (%) |
| | 2 | n (%) | n (%) | n (%) | n (%) |
| | >=3 | n (%) | n (%) | n (%) | n (%) |
| Day 21 | Arm for Infusion | | | | |
| J | | n (%) | n (%) | n (%) | n (%) |
| | Full Infusion Given | | | | |
| | | n (%) | n (%) | n (%) | n (%) |


| | Infusion Interrupted | n (%) | n (%) | n (%) | n (%) |
|---|---|---|---|---|---|
| Day 49 | Arm for Infusion | n (%) | n (%) | n (%) | n (%) |
| | Full Infusion Given | n (%) | n (%) | n (%) | n (%) |
| | Infusion Interrupted | n (%) | n (%) | n (%) | n (%) |
| Total Expo | osure (mL) | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx | XX, XX |

Note: N = Number of subjects in the Safety Population. n = Number of subjects in the specific category. Percentages are calculated as  $100 \times (n/N)$ . path\t\_program.sas date time

Table 14.2.8.1 Change in Total Polyp Score (TPS) from Baseline to Week 12 No Imputation MITT Population

| | | AK001 | AK001 | AK001 |
|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined [4] |
| Time Point | (N=) | (N= ) | (N=) | (N=) |
| Baseline [1] | | | | |
| n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 12 | | | | |
| n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Change from Baseline to Week 12 | | | | |
| n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| LS Mean | xx.x <sup>[2]</sup> | XX.X <sup>[2]</sup> | xx.x <sup>[2]</sup> | xx.x [4] |
| 95% CI | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[4]}$ |
| LS Mean Difference (AK001 vs. Placebo) | | xx.x [3] | xx.x <sup>[3]</sup> | xx.x <sup>[4]</sup> |
| 95% CI | | $(xx, xx)^{[3]}$ | $(xx, xx)^{[3]}$ | $(xx, xx)^{[4]}$ |
| p-value | | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[4]</sup> |

### Overall 3-group ANOVA

#### Combined Treatment 2-group ANOVA

| Effect | DF <sup>[2]</sup> | SE [2] | Statistics [2] | p-value [2] | DF [4] | SE [4] | Statistics [4] | p-value [4] |
|---|---|---|---|---|---|---|---|---|
| Treatment | nn | xx.xx | xx.xx | 0.xxxx | nn | XX.XX | xx.xx | 0.xxxx |
| Baseline TPS | nn | xx.xx | XX.XX | 0.xxxx | nn | xx.xx | xx.xx | 0.xxxx |
| Asthma | nn | XX.XX | XX.XX | 0.xxxx | nn | XX.XX | XX.XX | 0.xxxx |

path\t program.sas date time

Programming note: Repeat table 14.2.8.2 for Imputation method: Missing values are imputed by the average value of the placebo group at each specific time point. Repeat table 14.2.8.3 for no imputation and ITT population

Repeat table 14.2.8.4 for no imputation and PP population

Baseline is defined as the last non-missing value prior to first dose of study drug.

[2] LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment and asthma status (stratification factor). Baseline TPS score was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.
[4] This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). No imputations are made for missing data.

Table 14.2.9.1 Change in Total Polyp Score (TPS) from Baseline over Time No Imputation MITT Population

| 25 mg (N= ) n xx.x (xx.xx) xx.x xx.x, xx.x | 250 mg (N=) n xx.x (xx.xx) xx.x xx.x, xx.x | Combined [4] (N=) n xx.x (xx.xx) xx.x xx.x n |
|---|---|---|
| n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x |
| xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x |
| xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x |
| xx.x<br>xx.x, xx.x | xx.x<br>xx.x, xx.x | XX.X<br>XX.X, XX.X |
| xx.x, xx.x | xx.x, xx.x<br>n | XX.X, XX.X |
| n | n | |
| | | n |
| | | n |
| xx.x (xx.xx) | ( | |
| | xx.x (xx.xx) | xx.x (xx.xx) |
| XX,X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| n | n | n |
| xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| xx.x <sup>[2]</sup> | xx.x <sup>[2]</sup> | xx.x <sup>[4]</sup> |
| $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[4]}$ |
| xx.x <sup>[3]</sup> | xx.x <sup>[3]</sup> | xx.x <sup>[4]</sup> |
| | | $(xx, xx)^{[4]}$ |
| 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[4]</sup> |
| | xx.x<br>xx.x, xx.x<br>n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x<br>xx.x, xx.x | xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx. |

| Overall 3-group | ANOVA | | | | Combined Treatment 2-group ANOVA | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | DF <sup>[2]</sup> | SE [2] | Statistics [2] | p-value [2] | <u>D</u> F <sup>[4]</sup> | SE [4] | Statistics [4] | p-value [4] |
| Treatment | nn | xx.xx | xx.xx | 0.xxxx | nn | xx.xx | XX.XX | 0.xxxx |
| Time | nn | XX.XX | xx.xx | 0.xxxx | nn | xx.xx | XX.XX | 0.xxxx |
| Treat*Time | nn | xx.xx | xx.xx | 0.xxxx | nn | xx.xx | XX.XX | 0.xxxx |
| Baseline TPS | nn | xx.xx | xx.xx | 0.xxxx | nn | xx.xx | XX.XX | 0.xxxx |
| Asthma | nn | xx.xx | xx.xx | 0.xxxx | nn | xx.xx | XX.XX | 0.xxxx |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t\_program.sas date time

Programming note: Table will include the following raw score visits: Baseline, Week 3, Week 7, and Week 16; and change from baseline for Week 3, Week 7, and Week 16. Repeat the following tables ---

Table 14.2.9.2 Change in Total Polyp Score (TPS) from Baseline over Time (With Imputation) (MITT Population)

Programming note: Please adda footnote for imputation method.

Table 14.2.9.3 Change in Total Polyp Score (TPS) from Baseline over Time (No Imputation) (ITT Population)

Table 14.2.9.4 Change in Total Polyp Score (TPS) from Baseline over Time (No Imputation) (PP Population)

Table 14.2.9.5 Change in Total Polyp Score (TPS) from Baseline over Time (No Imputation, No Interaction) (MITT Population)

Table 14.2.9.6 Percent Change in Total Polyp Score (TPS) from Baseline over Time (No Imputation, No Interaction) (MITT population)

Table 14.2.9.7 Absolute Measurements in Total Polyp Score (TPS) from Baseline over Time (No Imputation, No Interaction) (MITT population)

Programming note: Time factor will include baseline as a level but baseline will not be included as a covariate in the model (needs to be a footnote as well).

<sup>[2]</sup> LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction, and asthma status (stratification factor). Baseline TPS was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). No imputations are made for missing data.

**Table 14.2.9.8** Total Polyp Score (TPS) - Time to Response at Any Time **MITT Population** 

| | | AK001 | AK001 | AK001 |
|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined [4] |
| Response Criteria | (N=) | (N= ) | (N= ) | (N= ) |
| 1-point Reduction Response [1] | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) |
| Time to Response (days) | | | | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 25 <sup>th</sup> – 75 <sup>th</sup> Percentile | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| p-value | | $0.xxxx^{[2]}$ | $0.xxxx^{[2]}$ | 0.xxxx <sup>[4]</sup> |
| HR (95% CI) | | $xx.x (xx.x - xx.x)^{[3]}$ | $xx.x (xx.x - xx.x)^{[3]}$ | $xx.x (xx.x - xx.x)^{[}$ |
| p-value | | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[4]</sup> |

50% Reduction Response

path\t\_program.sas date time

Programming note: Table will include the following responses: 1-point Reduction, and 50% Reduction, where response is defined as 1-point, and 50% reduction in TPS score, respectively.

<sup>[1]</sup> Response is defined as 1-point or 50% reduction in TPS score. Any subject who does not provide an assessment at the specified time point for defining response will be considered to be a non-responder.

[2] p-value is from the log-rank test.

[3] HR, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a Cox PH model.

[4] Similar analysis as described above in [2] and [3] is performed for the combined AK001 groups vs. Placebo.

Table 14.2.10.1 Subgroup Analysis of TPS Score at Week 12 by Gender MITT Population

| Subgroup | Time Point | Placebo<br>(N=) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined [4]<br>(N= ) | p-value for<br>Gender Effect | p-value for Treatment<br>by Gender Interaction |
|---|---|---|---|---|---|---|---|
| Male | Change from Baseline <sup>[1]</sup> to Week 12 | | | | | 0.xxxx <sup>[5]</sup> | 0.xxxx <sup>[5]</sup> |
| | n | n | n | n | n | $0.xxxx^{[6]}$ | 0.xxxx [6] |
| | Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | | |
| | Median | XX.X | XX.X | XX.X | XX.X | | |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | | |
| | LS Mean | xx.x [2] | xx.x <sup>[2]</sup> | XX.X [2] | xx.x [4] | | |
| | 95% CI | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[4]}$ | | |
| | LS Mean Difference (AK001 – Placebo) | | xx.x [3] | xx.x <sup>[3]</sup> | xx.x [4] | | |
| | 95% CI | | $(xx, xx)^{[3]}$ | $(xx, xx)^{[3]}$ | $(xx, xx)^{[4]}$ | | |
| | p-value | | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[4]</sup> | | |
| Female | Change from Baseline <sup>[1]</sup> to Week 12 | | | | | | |
| | n | n | n | n | n | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | | |
| | Median | XX.X | XX.X | XX.X | XX.X | | |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | | |
| | LS Mean | xx.x [2] | xx.x <sup>[2]</sup> | XX.X [2] | XX.X [4] | | |
| | 95% CI | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[4]}$ | | |
| | LS Mean Difference (AK001 – Placebo) | | xx.x [3] | xx.x <sup>[3]</sup> | xx.x [4] | | |
| | 95% CI <sup>[2]</sup> | | $(xx, xx)^{[3]}$ | $(xx, xx)^{[3]}$ | (xx, xx) [4] | | |
| | p-value <sup>[2]</sup> | | 0.xxxx <sup>[3]</sup> | 0.xxxx [3] | 0.xxxx <sup>[4]</sup> | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

<sup>[2]</sup> LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment and asthma status (stratification factor). Baseline TPS score was included as a covariate. An unstructured covariance model was used.
[3] Results are from contrast statement in the model descirbed in footnote [2].

<sup>[4]</sup> This analysis is performed similar to the model described in footnote [2] (AK001 dose levels are combined into one group vs. placebo).

p-values are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, gender, treatment\*gender interaction, and asthma status (stratification factor). Baseline TPS score was included as a covariate. An unstructured covariance model was used. Should unstructured covariance model not coverge, compound symmetry will be used instead.

<sup>[6]</sup> This analysis is performed similar to the model described in footnote [5] (AK001 dose levels are combined into one group vs. placebo).

path\t program.sas date time

Programming note: Repeat this table for all subgroups as follows:

Table 14.2.10.2 for Subgroup Analysis of TPS Score at Week 12 by Age(< Median, ≥ Median)

Table 14.2.10.3 for Subgroup Analysis of TPS Score at Week 12 by Asthma (Yes, No)

Table 14.2.10.4 for Subgroup Analysis of TPS Score at Week 12 by 1-point reduction responder criteria

Table 14.2.10.5 for Subgroup Analysis of TPS Score at Week 12 by 20% reduction responder criteria

Table 14.2.10.6 for Subgroup Analysis of TPS Score at Week 12 by 30% reduction responder criteria

**Table 14.2.11** Change in Size of Polyps (Lund-Mackay Score) from Baseline to Week 12 **MITT Population** 

| Score Component | Time Point | Placebo<br>(N=) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined [4]<br>(N=) |
|---|---|---|---|---|---|
| Maxillary | Baseline [1] | | | | |
| <i>y</i> | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| | Week 12 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Change from Baseline to Week 12 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | LS Mean | xx.x <sup>[2]</sup> | xx.x <sup>[2]</sup> | xx.x <sup>[2]</sup> | xx.x <sup>[4]</sup> |
| | 95% CI | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[4]}$ |
| | LS Mean Difference (AK001 vs. Placebo) | | xx.x [3] | xx.x <sup>[3]</sup> | xx.x <sup>[4]</sup> |
| | 95% CI | | $(xx, xx)^{[3]}$ | $(xx, xx)^{[3]}$ | $(xx, xx)^{[4]}$ |
| | p-value | | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[4]</sup> |

Anterior Ethmoid

Baseline is defined as the last non-missing value prior to first dose of study drug.

[2] LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment and asthma status (stratification factor). Baseline Lund-Mackay score was included as a covariate. An unstructured covariance model was used.

[3] Results are from contrast statement in the model described above.

| [4] This analysis is performed similar to the model above (AK001 dose levels are combined int | o one group vs. placebo). |
|---|---|
|---|---|

path\t\_program.sas date time

Programming note: Table will include the following Lund-Mackay score components: Maxillary, Anterior ethmoid, Posterior ethmoid, Sphenoid, Frontal, Osteomeatal complex, and Total score.

# Table 14.2.12.1 Change in Peak Nasal Inspiration Flow (PNIF) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 3, Week 12 and Week 16; and change from baseline for Week 3, Week 12 and Week 16.

LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction, and asthma status (stratification factor). Baseline PNIF was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo).


### **Table 14.2.12.2** Peak Nasal Inspirational Flow (PNIF) - Time to Response at Any Time **MITT Population**

[1] Response is defined as 50% reduction in PNIF score. Any subject who does not provide an assessment at the specified time point for defining response will be considered to be a non-responder.

[2] p-value is from the log-rank test.
[3] HR, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a Cox PH model.
[4] Similar analysis as described above in [2] and [3] is performed for the combined AK001 groups vs. Placebo.

path\t\_program.sas date time

Programming note: This table is same as Table 14.2.9.8.

Table will include the following response: 50% Reduction, where response is defined as 50% reduction in PNIF score.

## Table 14.2.13.1 Change in Sense of Smell (UPSIT Total Score) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 2, Week 3, Week 7, Week 12 and Week 16. If feasible, repeat table by each odorant.

LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction, and asthma status (stratification factor). Baseline UPSIT score was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). Missing data was assumed to be a wrong response and no imputation was performed to replace.


### **Table 14.2.13.2** Sense of Smell (UPSIT) - Time to Response at Any Time **MITT Population**

[1] Response is defined as 50% reduction in UPSIT score. Any subject who does not provide an assessment at the specified time point for defining response will be considered to be a non-responder.

[2] p-value is from the log-rank test.
[3] HR, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a Cox PH model.
[4] Similar analysis as described above in [2] and [3] is performed for the combined AK001 groups vs. Placebo.

path\t\_program.sas date time

Programming note: This table is same as Table 14.2.9.8.

Table will include the following response: 50% Reduction, where response is defined as 50% reduction in UPSIT score.

Table 14.2.14.1 Sino-nasal Outcome Test-22 (SNOT-22) (Five Most Important Items) at Week 12 MITT Population

| | Placebo | AK001<br>25 mg | AK001<br>250 mg | AK001<br>Combined |
|---|---|---|---|---|
| Item | (N=) | (N= ) | (N=) | (N=) |
| Need to blow nose | n (%) [1] | n (%) | n (%) | n (%) |
| Nasal blockage | n (%) | n (%) | n (%) | n (%) |
| Sneezing | n (%) | n (%) | n (%) | n (%) |
| Runny nose | n (%) | n (%) | n (%) | n (%) |
| Cough | n (%) | n (%) | n (%) | n (%) |
| Post-nasal discharge | n (%) | n (%) | n (%) | n (%) |
| Thick nasal discharge | n (%) | n (%) | n (%) | n (%) |
| Ear fullness | n (%) | n (%) | n (%) | n (%) |
| Dizziness | n (%) | n (%) | n (%) | n (%) |
| Ear pain | n (%) | n (%) | n (%) | n (%) |
| Facial pain/pressure | n (%) | n (%) | n (%) | n (%) |

Number (%) are based on the number of subjects that have picked the category as one of the five most important items. Missing data was imputed by the average score of the items present.

path\t\_program.sas date time

Programming note: Table will include all 22 items in Appendix F.


# Table 14.2.14.2 Change in SNOT-22 (Total Score of Five Most Important Items) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 2, Week 3, Week 7, Week 12 and Week 16.

LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction, and asthma status (stratification factor). Baseline SNOT-22 score was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). Missing data was imputed by the average score of the items present.

## Table 14.2.14.3 Change in SNOT-22 (Total Score of All Items) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

[3] Results are from contrast statement in the model described above.

[4] This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). Missing data was imputed by the average score of the items present.

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 2, Week 3, Week 7, Week 12 and Week 16.


LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction, and asthma status (stratification factor). Baseline SNOT-22 score was included as a covariate. An unstructured covariance model was used.


### **Table 14.2.14.4** Sino-nasal Outcome Test-22 (SNOT-22) – Time to Response at Any Time **MITT Population**

[1] Response is defined as 50% reduction in SNOT-22 score. Any subject who does not provide an assessment at the specified time point for defining response will be considered to be a non-responder.

[2] p-value is from the log-rank test.
[3] HR, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a Cox PH model.
[4] Similar analysis as described above in [2] and [3] is performed for the combined AK001 groups vs. Placebo.

path\t\_program.sas date time

Programming note: This table is same as Table 14.2.9.8.

Table will include the following response: 50% Reduction, where response is defined as 50% reduction in SNOT-22 score.

**Table 14.2.15.1** Visual Analogue Scale (VAS) by Symptom **MITT Population** 

| Symptom | Severity | Time Point | Placebo<br>(N=) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N=) | AK001<br>Combined<br>(N=) |
|---|---|---|---|---|---|---|
| Anterior Nasal Discharge | Mild <sup>[2]</sup> | Baseline [1]<br>Week 12 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| | Moderate <sup>[2]</sup> | Baseline [1]<br>Week 12 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| | Severe <sup>[2]</sup> | Baseline [1]<br>Week 12 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |

Posterior Nasal Discharge

path\t\_program.sas date time

Programming note: Table will include the following symptoms of rhinosinusitis: Anterior nasal discharge, Posterior nasal discharge, Nasal congestion, blockade, or obstruction, Decreased sense of smell, Facial pain or pressure.

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.
[2] The symptomatology can be divided into "mild", "moderate", and "severe" categories based on total score: Mild=0,1,2; Moderate=3,4,5,6; Severe=7,8,9,10 Missing data was imputed by the average score of the non-missing values.

Table 14.2.15.2 Change in Visual Analogue Scale (VAS by Symptom) from Baseline over Time MITT Population

| Symptom | Time Point | Placebo<br>(N=) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N=) | AK001<br>Combined [4]<br>(N=) |
|---|---|---|---|---|---|
| Anterior Nasal Discharg | e Baseline [1] | | | | |
| Anterior Musur Disenting | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| | Week 12 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| | Change from Baseline to Week 12 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | LS Mean | xx.x <sup>[2]</sup> | xx.x <sup>[2]</sup> | xx.x <sup>[2]</sup> | xx.x <sup>[4]</sup> |
| | 95% CI | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[2]}$ | $(xx, xx)^{[4]}$ |
| | LS Mean Difference (AK001 vs. Placebo) | | xx.x [3] | xx.x [3] | xx.x <sup>[4]</sup> |
| | 95% CI | | $(xx, xx)^{[3]}$ | $(xx, xx)^{[3]}$ | $(xx, xx)^{[4]}$ |
| | p-value | | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[3]</sup> | 0.xxxx <sup>[4]</sup> |

Posterior Nasal Discharge

. . .

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

<sup>[2]</sup> LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction and asthma status (stratification factor). Baseline VAS score was included as a covariate. An unstructured covariance model was used.

path\t program.sas date time

Programming note: Table will include the following symptom of rhinosinusitis: Anterior nasal discharge, Posterior nasal discharge, Nasal congestion, blockade, or obstruction, Decreased sense of smell, and Facial pain or pressure.

Programming note: Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 2, Week 3, Week 7, Week 12 and Week 16.

<sup>[3]</sup> Results are from contrast statement in the model described above.
[4] This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). Missing data was imputed by the average score of the non-missing values.

### Table 14.2.15.3 Change in Visual Analogue Scale (VAS Total Score) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 2, Week 3, Week 7, Week 12 and Week 16.

LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction and asthma status (stratification factor). Baseline VAS score was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). Missing data was imputed by the average score of the non-missing values.


### **Table 14.2.15.4** Visual Analogue Scale (VAS) – Time to Response at Any Time **MITT Population**

[1] Response is defined as 50% reduction in VAS score. Any subject who does not provide an assessment at the specified time point for defining response will be considered to be a non-responder.

[2] p-value is from the log-rank test.
[3] HR, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a Cox PH model.
[4] Similar analysis as described above in [2] and [3] is performed for the combined AK001 groups vs. Placebo.

path\t\_program.sas date time

Programming note: This table is same as Table 14.2.9.8.

Table will include the following response: 50% Reduction, where response is defined as 50% reduction in VAS score.

# Table 14.2.15.5 Change in Clinical Symptoms Improvement Scale (Total Score) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

[3] Results are from contrast statement in the model described above.

[4] This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo).

In case of Visit-Baseline, negative difference means improvement.

Missing data was imputed by the average score of the non-missing values.

path\t program.sas date tim

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 2, Week 3, Week 7, Week 12 and Week 16.


LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction and asthma status (stratification factor). Baseline Clinical Symptoms Improvement Scale score was included as a covariate. An unstructured covariance model was used.

# Table 14.2.16 Change in 36-Item Short Form Health Survey (SF-36 Total Score) from Baseline over Time MITT Population

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 3, Week 7, Week 12 and Week 16; and change from baseline for Week 3, Week 7, Week 12 and Week 16.

LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction and asthma status (stratification factor). Baseline SF-36 score was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo). Missing data was imputed by the average score of the category that the question belongs to.

# Table 14.2.17.1 Biomarker Analysis: Change in Biomarkers from Baseline over Time Biomarker Population, Sub-Study

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

Footnote: The content of this table is only a placeholder until we see the Biomarker test data

path\t program.sas date time

Programming note: This table is same as Table 14.2.9.1.

Table will include the following raw score visits: Baseline, Week 2, Week 3, Week 7, and Week 16; and change from baseline for Week 2, Week 3, Week 7, and Week 16. Table will include the following biomarkers: Eosinophilic Cationic Protein(µg/L), Histamin (ng/mL), Tryptase(ng/mL), Prostaglandins(pg/mL), Leukotrienes(pg/mL), Chymase(ng/mL), Carboxypeptidase A3(mg), Cytokines(mg), Chemokines (including Interleukin-5(ng/mL), Interleukin-17(ng/mL), Interleukin-17(ng/mL), Interleukin-13(ng/mL), Thymic Stromal Lymphopoietin(ng/mL), Interleukin-33(ng/mL), Interleukin-8(ng/mL)), Tumor Necrosis Factor(ng/mL), Albumin(µg/dL), Myeloperoxidase(unit/mL), Growth Factors.

Repeat Table 14.2.17.2 for Biomarker Analysis: Percent Change in Biomarkers from Baseline over Time (Biomarker Population, Sub-Study)
Repeat Table 14.2.17.3 for Biomarker Analysis: Change in Biomarkers from Baseline over Time (Biomarker Population, All Patients)
Repeat Table 14.2.17.4 for Biomarker Analysis: Percent Change in Biomarkers from Baseline over Time (Biomarker Population, All Patients)
Programming note: Tables 14.2.17.3 and 14.2.17.4 will include the following raw score visits: Baseline, Week 3, Week 7 and Week 12; and change from baseline for Week 3, Week 7 and Week 12. Tables 14.2.17.3 and 14.2.17.4 will include the following inflammatory responses: Eosinophils (10°/L), Mast Cells (10°/L), Basophils (10°/L).

<sup>[2]</sup> LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment, time, treatment\*time interaction, and asthma status (stratification factor). Baseline Biomarker level was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo).

Allakos, Inc.
AK001-002

#### Table 14.2.18.1 Change in Forced Expiratory Volume in 1 Second (FEV1) from Baseline to Week 7 MITT Population in Patients with Comorbid Asthma

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: This table is same as Table 14.2.8.1. Programming note: do not include asthma as a covariate. Programming note: Repeat the following tables ---

rogramming note: Repeat the joilowing tables ---Table 14.2.18.2 Change in Forced Vital Capacity (FVC) from Baseline to Week 7

Table 14.2.18.2 Change in Forced Vital Capacity (FVC) from Baseline to Week / Table 14.2.18.3 Change in Forced Expiratory Flow (FEF) from Baseline to Week 7 Table 14.2.18.4 Change in Asthma Control Test (ACT) from Baseline to Week 12

<sup>&</sup>lt;sup>[2]</sup> LS means, 95% CIs, and p-values comparing AK001 treatment groups to placebo group are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for treatment. Baseline FEV1 was included as a covariate. An unstructured covariance model was used.

<sup>[3]</sup> Results are from contrast statement in the model described above.

<sup>[4]</sup> This analysis is performed similar to the model above (AK001 dose levels are combined into one group vs. placebo).

Table 14.2.18.5.1
Use of Asthma Rescue Therapy<sup>[1]</sup> from Baseline to Week 12
MITT Population in Patients with Comorbid Asthma

| Time Point | Placebo<br>(N=) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N=) | AK001<br>Combined<br>(N=) |
|---|---|---|---|---|
| Baseline [2] | | | | |
| Daily user | n (%) | n (%) | n (%) | n (%) |
| Weekly user | n (%) | n (%) | n (%) | n (%) |
| Non-user | n (%) | n (%) | n (%) | n (%) |
| Veek 12 | | | | |
| Daily user | n (%) | n (%) | n (%) | n (%) |
| Weekly user | n (%) | n (%) | n (%) | n (%) |
| Non-user | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Question ACT4 from the ACT questionnaire. Daily User (3 or more times per day); Weekly User (2 or 3 times per week; once a week or less); Non-User (Not at all).

<sup>&</sup>lt;sup>[2]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Table 14.2.18.5.2
Use of Asthma Rescue Therapy<sup>[1]</sup> – Shift from Baseline to Week 12
MITT Population in Patients with Comorbid Asthma

| | Placebo (N= ) Baseline [2] | | | | | 25<br>(N | (001<br>mg<br>= )<br>line [2] | | | 25<br>(1 | K001<br>0 mg<br>N= )<br>eline [2] | AK001<br>Combined<br>(N= )<br>Baseline <sup>[2</sup> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Visit | Daily<br>user | Weekly<br>user | | Missing | Daily<br>user | Weekly<br>user | Non-user | Missing | Daily<br>user | Weekly<br>user | Non-user | Missing | Daily<br>user | Weekly<br>user | | Missing |
| Week 12 | | | | | | | | | | | | | | | | |
| Daily user | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| , | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Weekly user | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| , | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Non-user | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Question ACT4 from the ACT questionnaire . Daily User (3 or more times per day; 1 or 2 times per day); Weekly User (2 or 3 times per week; once a week or less); Non-User (Not at all).

Baseline is defined as the last non-missing value prior to first dose of study drug.

Table 14.3.1.19.1 Overall Summary of All Adverse Events Safety Population

| | D1 1 | AK001 | AK001 | AK001 |
|---|---|---|---|---|
| | Placebo | 25 mg | 250 mg | Combined |
| | (N=) | (N= ) | (N= ) | (N= ) |
| Subjetcs with any AE | n (%) | n (%) | n (%) | n (%) |
| Aubjects with any non-TEAE | n(%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE | n (%) | n (%) | n (%) | n (%) |
| Subjects with any Severe TEAE | n (%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE Related to Study Drug [1] | n (%) | n (%) | n (%) | n (%) |
| Subjects with any Serious TEAE | n (%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE with Outcome of Death | n (%) | n (%) | n (%) | n (%) |
| Subjects with any Treatment-Emergent AESI | n (%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE Leading to Dose Reduction | n (%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE Leading to Dose Interruption | n (%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE Leading to Study Drug Withdrawal | n (%) | n (%) | n (%) | n (%) |
| Subjects with any TEAE Leading to Dose Reduction, Interruption, or Withdrawal | n (%) | n (%) | n (%) | n (%) |
| Total Number of TEAE | n | n | n | n |
| Total Number of Severe TEAE | n | n | n | n |
| Γotal Number of TEAE Related to Study Drug [1] | n | n | n | n |
| Total Number of Serious TEAE | n | n | n | n |
| Total Number of TEAE with Outcome of Death | n | n | n | n |
| Total Number of TEAE Leading to Dose Reduction | n | n | n | n |
| Total Number of TEAE Leading to Dose Interruption | n | n | n | n |
| Total Number of TEAE Leading to Study Drug Withdrawal | n | n | n | n |
| Total Number of TEAE Leading to Dose Reduction, Interruption, or Withdrawal | n | n | n | n |

<sup>[1]</sup> Includes all events reported as "Possibly Related" or "Related" to study drug.

Table 14.3.1.19.2.1
Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
Safety Population

| System Organ Class / | Place<br>(N= | bo<br>) | AK0<br>25 m<br>(N= | | AK00<br>250 n<br>(N= | ng | AK0<br>Combi<br>(N= | ined |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

Table 14.3.1.19.2.2
Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Severity Safety Population

| System Organ Class / | Placebo<br>(N= ) | | | AK001<br>25 mg<br>(N= ) | | | AK001<br>250 mg<br>(N= ) | | | | AK001<br>Combined<br>(N= ) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Mild | Moderate | Severe | Missing | Mild | Moderate | Severe | Missing | Mild | Moderate | Severe | Missing | Mild | Moderate | Severe | Missing |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ·<br>· | | | | | | | | | | | | | | | | |
| System Organ Class 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| . To be continued on Page 2 for "All Active AK00." | I" aroun | | | | | | | | | | | | | | | |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the worst severity. path\t\_program.sas date time

Table 14.3.1.19.2.3 Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Relationship to Study Drug **Safety Population** 

| System Organ Class / | Placebo<br>(N= ) | | | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | | Cor<br>(! | K001<br>mbined<br>N= ) |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | Related [1] | Not Related [2] | Related [1] | Not Related [2] | Related [1] | Not Related [2] | Related [1] | Not Related [2] |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1<br>Preferred Term 1<br>Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| • | | | | | | | | |
| System Organ Class 2<br>Preferred Term 1<br>Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the strongest relationship to study drug.

[1] Includes all events reported by the Investigator as "Possibly Related," or "Related" to study drug.

[2] Includes all events reported by the Investigator as "Unlikely Related" or "Not Related" to study drug.

path\t program.sas date time

Table 14.3.2.19.3
Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term Safety Population

| System Organ Class / | Place<br>(N= | | AK00<br>25 m<br>(N= | | AK00<br>250 n<br>(N= | | AK001<br>Combined<br>(N= ) | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

Programming note: Repeat table for the tables listed below

Table 14.3.2.19.4.1 Treatment-Emergent Fatal Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)

Table 14.3.2.19.4.2 Treatment-Emergent Non-Fatal Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.19.5 Treatment-Emergent Severe Adverse Events by System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.19.6 Day 0 Treatment Emergent Adverse Events by System Organ Class and Preferred Term **Safety Population** 

| System Organ Class / | Placel<br>(N= | )<br>) | AK00<br>25 m<br>(N= | | AK00<br>250 r<br>(N= | ng | AK0<br>Comb<br>(N= | ined<br>) |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| S. story Oraco Class 2 | (0/) | | (0/) | | (0/) | | (0/) | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once. Note: Day-0 TEAEs, defined as all TEAEs occurring on the same calendar day as dosing (Day 0) with an onset on or after the time of the first dose of study drug.

Programming note: This table needs to be stand alone and every table after this one should be renumbered.

Post-Treatment Adverse Events by System Organ Class and Preferred Term **Safety Population** 

| System Organ Class / | Place | ho | AK0<br>25 n | | AK00<br>250 m | | AK(<br>Comb | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | (N= | ) | (N= | • | (N= | ) | (N= | |
| | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| • | | | | | | | | |
| • | | | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n | n (%) | n |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once. Note: Post-treatment adverse events are defined as TEAEs that have an onset more than 7 days after the last dose of study drug.

Programming note: Repeat table for the tables listed below

| Table 14.3.1.19.8.1 | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety Population Subgroup: Asthma Present) |
|---|---|
| Table 14.3.1.19.8.2 | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety Population Subgroup: Asthma Absent) |
| Table 14.3.1.19.8.3 | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety Population Subgroup: Using Concomitant Medication at Any Time During the |
| | Study) |
| Table 14.3.1.19.8.4 | Treatment-Emergent Adverse Events by SOC and Preferred Term (Safety Population Subgroup: Not Using Concomitant Medication at Any Time During the |
| | Study) |
| Table 14.3.1.19.8.5 | Treatment-Emergent Adverse Events by SOC and Preferred Term in at least 5 Subjects in any of Treatment Group (Safety Population) |


Table 14.3.4.20.1.1 Hematology Values and Changes from Baseline at All Visits – Conventional Units Safety Population

| Laboratory Parameter | Target Visit | Placebo<br>(N= ) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) |
|---|---|---|---|---|---|
| WBC (10 <sup>9</sup> /L) | Baseline [1] | | | | |
| WBC (10 /L) | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| | Week 2 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Change from Baseline to Week 2 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Neutrophils (10 <sup>9</sup> /L) | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug. path\t program.sas date time

Programming note: Table will include all hematology parameters collected from Central Laboratory, and all target visits (Week 2, Week 3, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Repeat for Table 14.3.4.20.1.2 using SI Units.

Table 14.3.4.20.1.3 Hematology – Shift from Baseline Safety Population

| | | | (1) | acebo<br>N= )<br>eline <sup>[1]</sup> | | AK001<br>25 mg<br>(N= )<br>Baseline [1] | | | | | AK<br>250<br>(N=<br>Basel | mg<br>= ) | | AK001<br>Combined<br>(N= )<br>Baseline [1] | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter | Target Visit | Low | Norma | l High | Missing | Low | Normal | High | Missing | Low | Normal | High | Missing | Low | Normal | High | Missing |
| WBC | Week 2 | | | | | | | | | | | | | | | | |
| | Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Week 3 | | | | | | | | | | | | | | | | |
| | Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Neutrophils | | | | | | | | | | | | | | | | | |
| ••• | | | | | | | | | | | | | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Programming note: Table will include all hematology parameters collected from Central Laboratory and all target visits (Week 2, Week 3, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Table 14.3.4.20.2.1
Serum Chemistry Values and Changes from Baseline at All Visits – Conventional Units
Safety Population

| Laboratory Parameter | Target Visit | Placebo<br>(N= ) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) |
|---|---|---|---|---|---|
| ALT (SGPT) (U/L) | Baseline [1] | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |
| | Week 2 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Change from Baseline to Week 2 | | | | |
| | n | n | n | n | n |
| | Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| AST (SGOT) (U/L) | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Programming note: Table will include all serum chemistry parameters collected by Central Laboratory and all target visits (Week 2, Week 3, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Repeat for Table 14.3.4.20.2.2 using SI Units.

Table 14.3.4.20.2.3 Serum Chemistry – Shift from Baseline Safety Population

| | Placebo<br>(N= )<br>Baseline [1] | | | AK001<br>25 mg<br>(N= )<br>Baseline [1] | | | AK001<br>250 mg<br>(N= )<br>Baseline [1] | | | AK001<br>Combined<br>(N= )<br>Baseline [1] | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter | Target Visit | Low | Normal | High | Missing | Low | Normal | High | Missing | Low | Normal | High | Missing | Low | Normal | High | Missing |
| ALT(SGPT) | Week 2 | | | | | | | | | | | | | | | | |
| | Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Week 3 | | | | | | | | | | | | | | | | |
| | Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AST (SGOT) | | | | | | | | | | | | | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Programming note: Table will include all serum chemistry parameters collected by Central Laboratory and all target visits (Week 2, Week 3, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Missing category was present.

Table 14.3.4.20.3.1 Urinalysis Values at All Visits Safety Population

| | Placebo | AK001<br>25 mg | AK001<br>250 mg | AK001<br>Combined |
|---|---|---|---|---|
| Target Visit | (N= ) | (N= ) | (N= ) | (N= ) |
| Densition [II] | | | | |
| | | | | n |
| | | | | xx.x (xx.xx) |
| | | | | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 2 | | | | |
| n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Change from Baseline to Week 2 | | | | |
| n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | XX.X | XX.X | xx.x | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | , | , | , | , |
| ••• | | | | |
| | Baseline [1] n Mean (SD) Median Min, Max Week 2 n Mean (SD) Median Min, Max Change from Baseline to Week 2 n Mean (SD) Median Min, Max | Baseline [1] n | Placebo | Placebo |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Programming note: Table will include pH and specific gravity using descriptive statistics at baseline and at each post-baseline time point for all target visits (Week 2, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

| Table will also include Categorical Laboratory Parameters, summarized by trea Instead of mean, median, min, max, use the lab reported values (for example, 0, displayed in the table. | atment group for each target week using counts are trace, $+1$ , $+2$ , etc). For these categorical laborat | nd percent of subjects in each result category.<br>ory parameters, no change from baseline will be |
|---|---|---|
| ak001-002_statistical analysis plan_final_v1_2017_08_16 | | CONFIDENTIAL |

### Table 14.3.4.20.3.2.1 Urinalysis – Shift from Baseline Part 1 of 2 Safety Population

| | | | (1) | acebo<br>N= )<br>eline [1] | | | 25<br>(N | 1001<br>mg<br>= )<br>line [1] | | | 25<br>(1 | K001<br>60 mg<br>N= )<br>eline [1] | | | Com<br>(N: | 001<br>bined<br>= )<br>line [1] | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter | Target Visit | Low | Normal | High | Missing | Low | Normal | High | Missing | Low | Normal | High | Missing | Low | Normal | High | Missing |
| РН | Week 2 | | | | | | | | | | | | | | | | |
| | Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Week 7 | | | | | | | | | | | | | | | | |
| | Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | ••• | | | | | | | | | | | | | | | | |
| Specific Gravity | | | | | | | | | | | | | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t\_program.sas date time

Programming note: Table will include only pH and specific gravity collected by Central Laboratory and all target visits (Week 2, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

#### Table 14.3.4.20.3.2.2 Urinalysis – Shift from Baseline Part 2 of 2 Safety Population

| | | Placebo<br>(N= )<br>Baseline [1] | | | AK001<br>25 mg<br>(N= )<br>Baseline [1] | | | AK001<br>250 mg<br>(N= )<br>Baseline [1] | | | AK001<br>Combined<br>(N= )<br>Baseline [1] | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Parameter | Target Visit | Negative | Positive | Missing | Negative | Positive | Missing | Negative | Positive | Missing | Negative | Positive | Missing |
| Blood | Week 2 | | | | | | | | | | | | |
| | Negative | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Positive | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Week 7 | | | | | | | | | | | | |
| | Negative | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Positive | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | Missing | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | ••• | | | | | | | | | | | | |
| Ketones | | | | | | | | | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t\_program.sas date time

Programming note: Table will include categorical laboratory parameters collected by Central Laboratory and all target visits (Week 2, Week 7, Week 12, and Week 16) and for Last Available On-Treatment Value. Please see Appendix A for visit windows. Instead of low, normal, high, use negative, positive categories.

Table 14.3.4.21.1 Vital Signs - Day 0 Pre-Dose and Post-Dose Safety Population

| Vital Sign | Time Point | Placebo<br>(N= ) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) |
|---|---|---|---|---|---|
| Systolic BP (mmHg) | Day 0 Pre-Dose [1] n Mean (SD) Median Min, Max | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x |
| | Day 0 Post-Dose [2] Change from Baseline to Day 0 Post-Dose | | | | |
| Diastolic BP (mmHg) | | | | | |

<sup>[1]</sup> Day 0 Pre-Dose is defined as the pre-dose value on Day 0. [2] Day 0 Post-Dose is approximately 15 min after post-dose.

Programming note: Table will include the following vital signs: systolic BP (mmHg), diastolic BP (mmHg), pulse rate (beats/min), body temperature (°C) and respiration rate (breaths/min).

Table 14.3.4.21.2
Vital Signs – Screening and Post Day 0
Safety Population

| Vital Sign | Target Visit | Placebo<br>(N= ) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) |
|---|---|---|---|---|---|
| Systolic BP (mmHg) | Screening n Mean (SD) Median Min, Max Baseline [1] | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | n<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| | Week 2 Change from Baseline to Week 2 | | | | |
| Diastolic BP (mmHg) | | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Programming note: Table will include the following vital signs: systolic BP (mmHg), diastolic BP (mmHg), pulse rate (beats/min), body temperature (°C) and respiration rate (breaths/min) for the following target visits: Screening, Baseline, Week 2, Week 3, Week 7, Week 12, and Week 16, and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Table 14.3.4.21.3
Incidence of Potentially Clinically Significant Vital Sign Results
Safety Population

| Any Post-Baseline<br>Clinically Significant Abnormalities? | Potentially Clinically<br>Significant Criteria | Target Visit | Placebo<br>(N= ) | AK001<br>25 mg<br>(N= ) | AK001<br>250 mg<br>(N= ) | AK001<br>Combined<br>(N= ) |
|---|---|---|---|---|---|---|
| Systolic Blood Pressure | Criteria | Baseline<br>Any Post-Baseline Visit<br>Day 0 Post-Dose<br>Week 2 | n (%)<br>n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%)<br>n (%) |
| Diastolic Blood Pressure | Criteria | Baseline Any Post-Baseline Visit Day 0 Post-Dose Week 2 | n (%)<br>n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%)<br>n (%) | n (%) n (%) n (%) n (%) n (%) | n (%)<br>n (%)<br>n (%)<br>n (%) |
| | | | 11 (70) | 11 (70) | 11 (70) | 11 (70) |

Programming note: Table will include all parameters (systolic BP (mmHg), diastolic BP (mmHg), pulse rate(beats/min), body temperature (°C) and respiration rate (breaths/min)) with defined potentially clinically significant ranges at each post-Baseline visit. Target visits for all parameters after Day 0 are: Week 2, Week 3, Week 7, Week 12, and Week 16. Please see Appendix A for visit windows.

## **Appendix J: Figure Layouts**


| Figure | Figure 14.2.1.1 |
|---|---|
| Title 1 | Least Squares Mean Change in Total Polyp Score (TPS) |
| Title 2 | MITT Population |
| Type of graph | Line Graph |
| y-axis | Mean Change in TPS |
| y-axis (label) | Least Squares Mean Change (95% CI) in TPS |
| x-axis | 3, 7, 12, 16 Weeks (programming note: time points will change with different efficacy outcomes) |
| x-axis (label) | Time Point |
| Legend | No. of patients |
| | AK001 25 mg n n n n |
| | AK001 250 mg n n n n |
| | AK001 Combined n n n n |
| | Placebo n n n n |
| Footnotes | Note: Bars represent 95% CIs. |
| | Figure corresponds to Table 9.1 |
| 4.11:: 1: 0 | path\t_program.sas date time |
| Additional information | Plot Least Squares Mean Change from Baseline and 95% CIs. |
| | Repeat Figure 14.2.1.2 – Mean Change in Total Polyp Score (TPS) (MITT Population in Patients with Cormobid Asthma) |
| | Repeat Figure 14.2.2 – Mean Change in Peak Nasal Inspiratory Flow (PNIF) (MITT Population) |
| | Repeat Figure 14.2.3 – Mean Change in University of Pennsylvania Smell Identification Test (UPSIT) (MITT Population) |

| Allakos, Inc. | Statistical Analysis Plan |
|---------------|---------------------------|
| AK001-002 | 16 August 2017 |

| Repeat Figure 14.2.4 – Mean Change in 22-item Sinonasal Outcome Test (SNOT-22) (MITT Population) |
|---|
| Repeat Figure 14.2.5 – Mean Change in Visual Analogue Scale (VAS) (MITT Population) |
| Repeat Figure 14.2.6 – Mean Change in Forced Expiratory Volume in 1 Second (FEV1) (MITT Population in Patients with Cormobid Asthma) |
| Repeat Figure 14.2.7 – Mean Change in Asthma Control Test (ACT) (MITT Population in Patients with Cormobid Asthma) |
| Repeat Figure 14.2.8 – Mean Change in Blood Eosinophil Count (Biomarker Population) |

Allakos, Inc.
AK001-002

| Figure | Figure 14.2.1 | Figure 14.2.1.3 | | | |
|---|---|---|---|---|---|
| Title 1 | Kaplan-Meier | Kaplan-Meier Curves for Time to 1-point Reduction in Total Polyp Score (TPS) | | | |
| Title 2 | | MITT Population | | | |
| Type of graph | Kaplan-Meier | Step Function | | | |
| y-axis | Survival Prob | ability | | | |
| y-axis (label) | Survival Prob | ability | | | |
| x-axis | Weeks | | | | |
| x-axis (label) | Survival Time | ( ) | | | |
| Legend | | AK001 25mg, Placebo | | | |
| Footnotes | Note: Figure | Note: Figure corresponds to Table 14.2.9.8 | | | |
| | .4.3. | | | | |
| A 111/2 12 0 /2 | path\t_progra | m.sas date | time | | |
| Additional information | D | | | 41 | |
| | Programming | g note: aaa a su <u>t</u><br>Placebo | | | of the cuves, as follon<br>AK001 Combined |
| | Median | xx.x | | AK001 250 mg | |
| | 95% CI | (xx.x, xx.x) | xx.x<br>(xx.x, xx.x) | xx.x<br>(xx.x, xx.x) | xx.x<br>(xx.x, xx.x) |
| | p-value | (лл.л, лл.л) | 0.xxxx | 0.xxxx | 0.xxxx |
| | HR | | xx.x | xx.x | xx.x |
| | 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | p-value | , , | 0.xxxx | 0.xxxx | 0.xxxx |

| Allakos, Inc. | Statistical Analysis Plan |
|---------------|---------------------------|
| AK001-002 | 16 August 2017 |


**Appendix K: Listing Layouts** 

**Listing 16.2.1.1.1 Subject Populations** 

| Subject | | ITT | Safety | MITT | PP | Biomarker |
|---|---|---|---|---|---|---|
| ID | Treatment Group | Population [1] | Population [2] | Population [3] | Population [4] | Population [5] |
| XXXXXX | XXXXXXXXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

Programming note: Sort by subject ID.

<sup>[1]</sup> All randomized subjects.
[2] All randomized subjects who take at least one dose of study drug.
[3] All randomized subjects who take at least one dose of the study drug and have both a baseline and at least one post-baseline efficacy assessment.
[4] All MITT population subjects who have a week 12 visit and valid efficacy measurements.
[5] All randomized subjects who has at least 1 sample obtained for biomarker analysis.

Listing 16.2.1.1.2 Subject Disposition

| a 1 | | | D | Reason for | a 1 1 | Date of Study | B () 4 ( 9.11 ( B)) |
|---|---|---|---|---|---|---|---|
| Subject | | Completed | Date of Last | Discontinuing | Completed | Completion / | Reason(s) that Subject Did |
| ID | Treatment Group | Treatment | Dose | Study Drug | Study | Discontinuation | Not Complete the Study |
| XXXXXX | XXXXXXXXX | Yes/No | Date | Reason | Yes/No | date9. | Reason* |
| XXXXXX | XXXXXXXXX | Yes/No | Date | Reason | Yes/No | date9. | Reason {including Other |
| | | | | | | | description} |
| XXXXXX | XXXXXXXXX | Yes/No | Date | Reason | Yes/No | date9. | Reason |
| XXXXXX | XXXXXXXXX | Yes/No | Date | Reason | Yes/No | date9. | Reason |
| XXXXXX | xxxxxxxxx | Yes/No | Date | Reason | Yes/No | date9. | Reason |

Note: \* indicates primary reason.

path\l\_program.sas date time

Programming note: Sort by subject ID.

Listing 16.2.1.1.3 Subject Visit Dates

| Subject ID | Treatment Group | Visit | Visit Date |
|------------|-----------------|-----------------|------------|
| | | | _ |
| XXXXXX | XXXXXXXXX | Screening | date |
| | | Baseline | |
| | | Day 0 | |
| | | Week 2 | |
| | | Week xx | |
| | | Week xx | |
| | | ••• | |
| | | Follow-up Visit | |
| | | Unscheduled | |
| XXXXXX | XXXXXXXXX | | |

Programming note: Sort by subject ID and visit date.

Listing 16.2.2.2 Protocol Deviations

| Subject ID | Treatment Group | Protocol Deviation<br>Category | Protocol Deviation<br>Type | Deviation Date | Deviation Time | Action Taken |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | category | type | date9. | time5. | action |
| | | | | date9. | time5. | action |
| XXXXXX | XXXXXXXXX | category | type | | | |
| XXXXXX | XXXXXXXXX | category | type | date9. | time5. | action |
| XXXXXX | XXXXXXXXX | category | type | date9. | time5. | action |

path\l program.sas date

time

Programming note: Sort by subject ID.

Programming note: Protocol Deviation Category includes Informed Consent, Randomization Error, Safety, Efficacy, IP/Treatment Deviation, and Other Protocol Deviations.

Protocol deviation Type includes Informed Consent Procedures and etc which was described on CRF form.

Listing 16.2.2.3 Inclusion/Exclusion Findings

| Subject<br>ID | Treatment Group | Meet All Eligibility<br>Criteria | If Re-Screen, Initial Screening Number | Criterion Type | Criterion No. | Protocol<br>Version Date |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXXXXXX | Yes/No | XXXXXX | Inclusion/Exclusion | XX | date9. |
| XXXXX | XXXXXXXXX | Yes/No | xxxxxx | Inclusion/Exclusion | XX | date9. |
| XXXXX | XXXXXXXXX | Yes/No | xxxxxx | Inclusion/Exclusion | XX | date9. |
| XXXXX | XXXXXXXXX | Yes/No | xxxxxx | Inclusion/Exclusion | XX | date9. |

Programming note: Sort by subject ID.

Listing 16.2.1.4.1 Informed Consent

| Subject Treatment<br>ID Group | Date Signed Informed<br>Consent | Protocol Version Date at<br>Initial Consent |
|---|---|---|
| xxxxxx xxxxxxxxx | date9. | xxxxxx |
| xxxxxx xxxxxxxxx | date9. | xxxxxx |
| xxxxxx xxxxxxxxx | date9. | xxxxxx |
| xxxxxx xxxxxxxxx | date9. | xxxxxx |
| | ••• | |

Programming note: Sort by subject ID and informed consent date, in the event of multiple forms. Programming note: Date of the initial consent form will be reposted.

Listing 16.2.1.4.2 Withdrawal of Consent

| Subject Treatment<br>ID Group | Withdrew Consent | Study Participant | Withdrew Date |
|---|---|---|---|
| xxxxxx xxxxxxxxx | Yes/No | xxxxxx | date9. |
| xxxxxx xxxxxxxxx | Yes/No | xxxxxx | date9. |
| xxxxxx xxxxxxxxx | Yes/No | xxxxxx | date9. |
| xxxxxx xxxxxxxxx | Yes/No | xxxxxx | date9. |

Programming note: Sort by subject ID.

Listing 16.2.4.5.1
Demographics and Baseline Characteristics
Part 1 of 2

| | Treatment | | Age | | | |
|---|---|---|---|---|---|---|
| Subject ID | Group | Region | (years) [1] | Gender | Ethnicity | Race |
| xxxxxx | xxxxxxxxx | Region | XX | Male/Female | Ethnicity | Race |
| XXXXXX | XXXXXXXXX | Region | XX | Male/Female | Ethnicity | Race |
| XXXXXX | XXXXXXXXX | Region | XX | Male/Female | Ethnicity | Race |
| XXXXXX | XXXXXXXXX | Region | XX | Male/Female | Ethnicity | Race |
| | | C | | | • | Race |
| | | | | | | Race |

[1] Age on Consent Date.

path\l\_program.sas date time

Listing 16.2.4.5.2
Demographics and Baseline Characteristics
Part 2 of 2

| Subject ID | Treatment<br>Group | Height (cm) | Weight (kg) | BMI (kg/m²) | TPS Score | Use of Asthma<br>Rescue Therapy |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXXXXXX | XX | XX | XX.X | XX.X | Yes/No |

Programming note: Sort by subject ID.
Listing 16.2.4.6
Relevant Respiratory Histroy at Screening

| | | | | Experienced | Had | | | If Yes, | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | Have | If Yes, | Asthma | Rhinosinusitus | | Have Aspirin | Diagnosis | |
| Subject ID | Group | Asthma? | Onset Date | Exacerbation? | Symptom? | If Yes, Symptom | Sensitivity? | Date | Ongoing? |
| XXXXXX | XXXXXXXXX | Yes/No | date9. | Yes/No | Yes/No | Anterior nasal discharge | Yes/No | date9. | Yes/No |
| XXXXXX | XXXXXXXXX | Yes/No | date9. | Yes/No | Yes/No | Posterior nasal discharge | Yes/No | date9. | Yes/No |
| XXXXXX | XXXXXXXXX | Yes/No | date9. | Yes/No | Yes/No | Decreased sense of smell | Yes/No | date9. | Yes/No |
| XXXXXX | xxxxxxxxx | Yes/No | date9. | Yes/No | Yes/No | Facial pain or pressure | Yes/No | date9. | Yes/No |
| | | | | | | • • | Yes/No | date9. | Yes/No |

path\l\_program.sas date time

Listing 16.2.4.7 Medical History at Screening

| Subject ID | Treatment Group | MedDRA System<br>Organ Class | Condition // MedDRA Preferred<br>Term | CRF Start/Stop Date<br>Unknown | Onset Date | Ongoing/Resolved | End Date |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | Body System | Verbatim term // MedDRA<br>Preferred Term | Checkbox | date9. | Ongoing/Resolved | date9. |
| | | Body System | Verbatim term // MedDRA Preferred Term | value | date9. | Ongoing/Resolved | date9. |
| | | Body System | Verbatim term // MedDRA<br>Preferred Term | | date9. | Ongoing/Resolved | date9. |
| xxxxxx | xxxxxxxxx | Body System | Verbatim term // MedDRA<br>Preferred Term | | date9. | Ongoing/Resolved | date9. |
| | | Body System | Verbatim term // MedDRA<br>Preferred Term | | date9. | Ongoing/Resolved | date9. |
| | | Body System | Verbatim term // MedDRA<br>Preferred Term | | date9. | Ongoing/Resolved | date9. |
| ••• | | | | | | | |

path\l\_program.sas date time

Programming note: sort by subject ID and onset date within each subject.

Listing 16.2.4.8 Physical and Neurological Examination

| Subject | Treatment | Target | Visit Date | | | Description of | |
|---|---|---|---|---|---|---|---|
| ID | Group | Visit | (Study Day) | Body System | Overall Assessment | Abnormality | Clinically Significant |
| VVVVV | VVVVVVVVVV | Screening | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| XXXXXX | XXXXXXXXX | Screening | dates. (xx) | | Normal/Abnormal | | Yes/No |
| | | | | Body System 2 | | Description | |
| | | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | | Day 1 Pre-Dose | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | Buy 1110 Bose | dutes. (AA) | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 2 Body System 3 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 5 | 1 vorman / romorman | Description | 1 03/110 |
| | | Day 1 Post-Dose | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | • | , | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | | | | | | • | |
| xxxxxx | xxxxxxxxx | Screening | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| ΛΛΛΛΛΛ | AAAAAAAAA | Screening | dates. (AA) | Body System 1 Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 2 Body System 3 | Normal/Abnormal | Description | Yes/No |
| | | | | Dody System 5 | Normal/Admornian | Description | 1 05/110 |
| | | Day 1 Pre-Dose | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | Ž | , | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | | Day 1 Post-Dose | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | | Body System 3 | Normal/Abnormal | Description | Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Listing 16.2.4.9 Symptom Directed Physical Examination

| Subject ID | Treatment<br>Group | Target Visit | Performed? | Exam Date<br>(Study Day) | Exam Time | Infusion Site Reaction? | New/Worsened CS findings? |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | Day 0 | Yes/No | date9. (xx) | time5. | Yes/No | Yes/No |
| | | Week 2 | Yes/No | date9. (xx) | time5. | Yes/No | Yes/No |
| | | Week 3 | Yes/No | date9. (xx) | time5. | Yes/No | Yes/No |
| XXXXXX | XXXXXXXXX | Day 0 | Yes/No | date9. (xx) | time5. | Yes/No | Yes/No |
| | | Week 2 | Yes/No | date9. (xx) | time5. | Yes/No | Yes/No |
| | | Week 3 | Yes/No | date9. (xx) | time5. | Yes/No | Yes/No |

. . .

Note: Study day is calculated as days since the date of first dose of study drug. CS=Clinically Significant

path\l\_program.sas date time

Listing 16.2.4.10 Electrocardiogram at Screening

| Subject<br>ID | Treatment Group | Performed? | Assessment<br>Date<br>(Study Day) | Assessment | Heart<br>Rate<br>(bpm) | PR<br>Interval<br>(ms) | RR<br>Interval<br>(ms) | QRS<br>Interval<br>(ms) | QT<br>Interval<br>(ms) | • | QTc Interval<br>(Bazett)<br>(ms) | Any Findings<br>Abnormal? <sup>[1]</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | Yes/No | date9. (xx) | time5. | xxx | xxx | xxx | xxx | xxx | xxx | xxx | Yes: CS/NCS /<br>No/cant/Unable to<br>evaluate |
| | | | date9. (xx) | time5. | xxx | xxx | xxx | xxx | xxx | XXX | xxx | evaluate |
| xxxxxx | xxxxxxxxx | Yes/No | date9. (xx)<br>date9. (xx) | time5.<br>time5. | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | |

Note: Study day is calculated as days since the date of first dose of study drug. CS=Clinically Significant; NCS=Not Clinically Significant [1] Investigator interpretation of ECG and clinical significance

path\l\_program.sas date time

Listing 16.2.4.11.1 Pregnancy Test

| | Treatment | | | If Yes, Type of | Reason if not | Test Date (Study | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Group | Visit | Performed? | Test | done | Day) | Test Time | Result |
| XXXXXX | XXXXXXXXX | Screening | Yes/No | Test | Surgically sterile | date9. (xx) | time5. | Negative/Positive |
| | | Day -3 | Yes/No | Test | Post-menopausal | date9. (xx) | time5. | Negative/Positive |
| | | Week x | Yes/No | Test | Other (Specify) | date9. (xx) | time5. | Negative/Positive |
| xxxxxx | xxxxxxxxx | Screening Day -3 Week x | Yes/No<br>Yes/No<br>Yes/No | Test<br>Test<br>Test | Surgically sterile<br>Post-menopausal<br>Other (Specify) | date9. (xx) | time5.<br>time5. | Negative/Positive<br>Negative/Positive<br>Negative/Positive |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Listing 16.2.4.11.2 Pregnancy Report during Study

| | | Patient or patient's | 3 | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | partner became | Pregnancy Date | Delivery | | Infant | Infant | Any Congenital |
| Subject ID | Group | pregnant? | (Study Day) | Date | Outcome | Weight (kg) | Height (cm) | Abnormalities? |
| XXXXXX | XXXXXXXXX | Yes/No | date9. (xx) | date9. | Normal/Abnormal | XX | XX | Yes/No |
| | | Yes/No | date9. (xx) | date9. | Normal/Abnormal | XX | XX | Yes/No |
| | | Yes/No | date9. (xx) | date9. | Normal/Abnormal | XX | XX | Yes/No |
| xxxxxx | xxxxxxxxx | Yes/No | date9. (xx) | date9. | Normal/Abnormal | XX | XX | Yes/No |
| | | Yes/No | date9. (xx) | date9. | Normal/Abnormal | XX | XX | Yes/No |
| | | Yes/No | date9. (xx) | date9. | Normal/Abnormal | XX | XX | Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Listing 16.2.4.12
Follicle-Stimulating Hormone (FSH) Test at Screening

| | Treatment | | Collection Date | Collection | |
|---|---|---|---|---|---|
| Subject ID | Group | Performed? | (Study Day) | Time | Result (IU/L) |
| xxxxxx | xxxxxxxxx | Yes/No | date9. (xx) | time5. | XX |
| | | Yes/No | date9. (xx) | time5. | XX |
| | | Yes/No | date9. (xx) | time5. | XX |
| XXXXXX | xxxxxxxxx | Yes/No | date9. (xx) | time5. | XX |
| | | Yes/No | date9. (xx) | time5. | XX |
| | | Yes/No | date9. (xx) | time5. | XX |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l program.sas date time

Programming note: Sort by subject ID.

Programming note:

Repeat Listing 16.2.4.13 for Fecal Sample Test at Screening {Replace column "Result (IU/L) with "Result", and display "Negative/Positive" in the result field}

Repeat Listing 16.2.4.14 for Anti-Drug Antibody (ADA) {Add a column "Target Visit" after "Treatment Group"; Replace column "Result (IU/L) with "Result"}

Repeat Listing 16.2.4.15 for Exploratory Biomarkers {Add a column "Target Visit" after "Treatment Group"; Replace column "Result (IU/L) with "Result", display all collected biomarkers analysis results}

Repeat Listing 16.2.4.16 for Serum Samples for Total Immunoglobulin E and ImmunoCAP on Day -3 {Add a column "Typet" after "Treatment Group"; Replace column "Result (IU/L) with "Result"}


Listing 16.2.4.17 Prior Medications

| Subject<br>ID | Treatment<br>Group | CM<br># | Verbatim Term //<br>Generic Name | Start Date<br>(Study Day) | Stop Date<br>(Study Day) | Dose | Units | Dose Form | Route | Frequency | Indication | Primary<br>Reason for<br>Medication |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term //<br>Generic Name | date9. (xx) | date9. (xx) | dose | unit | dose form | route | frequency | indication | xxxx |
| | | 2 | Verbatim Term // Generic Name | date9. (xx) | date9. (xx) | dose | unit | dose form | route | frequency | indication | xxxx |
| | | 3 | Verbatim Term //<br>Generic Name | date9. (xx) | date9. (xx) | dose | unit | dose form | route | frequency | indication | XXXX |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term //<br>Generic Name | date9. (xx) | date9. (xx) | dose | unit | dose form | route | frequency | indication | xxxx |
| | | 2 | Verbatim Term //<br>Generic Name | date9. (xx) | date9. (xx) | dose | unit | dose form | route | frequency | indication | xxxx |
| | | 3 | Verbatim Term //<br>Generic Name | date9. (xx) | date9. (xx) | dose | unit | dose form | route | frequency | indication | XXXX |

Note: Study day is calculated as days since the date of first dose of study drug. Prior Medications are those started within the 30 days before Screening.

path\l\_program.sas date time

Programming note: sort by subject ID and start date and stop date within each subject.

Programming note: Repeat listing 16.2.4.18 for Concomitant Medications {Replace prior footnote with "Concomitant medications are those medications taken at the start of study drug or initiated after the initial dose of study drug." Add a flag # for medication that start after the last dose of study drug.}

Listing 16.2.4.19 Intranasal Steroid Adjustment at Day 0

| Treatment | Completed | Start Data | End Data | |
|---|---|---|---|---|
| | | ~ | | |
| Group | Run-in? | (Study Day) | (Study Day) | Compliance (%) |
| xxxxxxxxx | Yes/No | date9. (xx) | date9. (xx) | XX.X |
| | Yes/No | date9. (xx) | date9. (xx) | XX.X |
| | Yes/No | date9. (xx) | date9. (xx) | XX.X |
| xxxxxxxxx | Yes/No | date9. (xx) | date9. (xx) | XX.X |
| | Yes/No | date9. (xx) | date9. (xx) | XX.X |
| | Yes/No | date9. (xx) | date9. (xx) | XX.X |
| | | Group Run-in? xxxxxxxxxx Yes/No Yes/No Yes/No xxxxxxxxxx Yes/No Yes/No | Group Run-in? (Study Day) xxxxxxxxxxx Yes/No date9. (xx) Yes/No date9. (xx) yes/No date9. (xx) xxxxxxxxxxx Yes/No date9. (xx) yes/No date9. (xx) | Group Run-in? (Study Day) (Study Day) xxxxxxxxxx Yes/No date9. (xx) date9. (xx) Yes/No date9. (xx) date9. (xx) Yes/No date9. (xx) date9. (xx) xxxxxxxxxx Yes/No date9. (xx) date9. (xx) Yes/No date9. (xx) date9. (xx) |

. . .

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

## Listing 16.2.5.20 Study Drug Administration

| Subject ID | Treatment<br>Group | Target<br>Visit | Drug<br>Administered? | Arm for Administration | Start Date | Start Time | End Time | Full Infusion<br>Given? | If Yes, Total<br>Volume (mL) | If No, Amount<br>Given | Infusion<br>Interrupted? | If Yes,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | Day 0 | Yes/No | Left/Right | date9. (xx) | time5. | time5. | Yes/No | XX | xx | Yes (#)/No | Reason |
| | | Week 3 | Yes/No | Left/Right | date9. (xx) | time5. | time5. | Yes/No | XX | XX | Yes (#)/No | Reason |
| | | Week 7 | Yes/No | Left/Right | date9. (xx) | time5. | time5. | Yes/No | XX | XX | Yes (#)/No | Reason |
| xxxxxx | xxxxxxxxx | Day 0 | Yes/No | Left/Right | date9. (xx) | time5. | time5. | Yes/No | XX | XX | Yes (#)/No | Reason |
| | | Week 3 | Yes/No | Left/Right | date9. (xx) | time5. | time5. | Yes/No | XX | XX | Yes (#)/No | Reason |
| | | Week 7 | Yes/No | Left/Right | date9. (xx) | time5. | time5. | Yes/No | XX | XX | Yes (#)/No | Reason |

. . .

Note: # is the number of times interrupted

path\l\_program.sas date time

Listing 16.2.6.21.1 Total Polyp Score (TPS)

| | Treatment | | | Date Performed | | |
|---|---|---|---|---|---|---|
| Subject ID | Group | Target Visit | Performed? | (Study Day) | Time | Total Score |
| XXXXXX | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | X |
| | | Baseline | Yes/No | date9. (xx) | time5. | X |
| | | Week X | Yes/No | date9. (xx) | time5. | X |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | X |
| | | Baseline | Yes/No | date9. (xx) | time5. | X |
| | | Week X | Yes/No | date9. (xx) | time5. | X |
| | | ••• | | | | |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

| Programming note | e: Repeat list | ing for the | listings listed below |
|------------------|----------------|-------------|-----------------------|
|------------------|----------------|-------------|-----------------------|

| Listing 16.2.6.21.2 | Size of Polyps (Lund-Mackay Score) {Add a column for "Lund-Mackay Scoring System" before |
|---|---|
| | "Total Score"} |
| Listing 16.2.6.21.3 | Peak Nasal Inspiratory Flow (PNIF) {Replace column "Total Score" with columns "Reading 1 |
| | (L/min)", "Reading 2 (L/min)", "Reading 3 (L/min)", "Highest Reading (L/min)"} |
| Listing 16.2.6.21.4 | University of Pennsylvania Smell Identification Test (UPSIT) |
| Listing 16.2.6.21.5 | Sino-nasal Outcome Test-22 (SNOT-22) {Add a column for "Five Most Important Items" before |
| | "Total Score", display items in the field} |
| Listing 16.2.6.21.6 | Visual Analogue Scale (VAS) {Add two columns for "Symptom" and "Severity"} |
| Listing 16.2.6.21.7 | Clinical Symptoms Improvement Scale |

Listing 16.2.6.21.8.1 36-Item Short Form Health Survey (SF-36) Part 1 of 3

| | Treatment | Target | | Date<br>Performed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | | Visit | | (Study Day) | Time | GH1 | HT | PF01 | PF02 | PF03 | PF04 | PF05 | PF06 | PF07 | PF08 | PF09 | PF10 |
| | - | | | | | | | | | | | | | | | | |
| XXXXXX | xxxxxxxxx | Day 0 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Week 3 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| xxxxxx | xxxxxxxxx | Day 0 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Week 3 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| xxxxxx | xxxxxxxxx | Day 0 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Week 3 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | | | | | | |
| xxxxxx | xxxxxxxxx | Day 0 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Week 3 | Yes/No | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| ••• | | | | | | | | | | | | | | | | | |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Programming note: Sort by subject ID.

Programming note: provide a key cover sheet for all the columns.

Listing 16.2.6.21.8.2 36-Item Short Form Health Survey (SF-36) Part 2 of 3

| Subject<br>ID | Treatment<br>Group | Target<br>Visit | RP1 | RP2 | RP3 | RP4 | RE1 | RE2 | RE3 | SF1 | RP1 | BP2 | VT1 | MH1 | MH2 | МН3 | VT2 | MH4 | VT3 | MH5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | огоцр | V 151t | 1(1 1 | 1012 | 1013 | 1(1 ) | TELL | TCD2 | TCLS | 51 1 | DI I | D1 2 | , , , , | 141111 | 141112 | 111113 | , 12 | 11111 | , 13 | |
| xxxxxx | xxxxxxxxx | Day 0 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Week 3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| XXXXXX | xxxxxxxxx | Day 0 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Week 3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| xxxxxx | xxxxxxxxx | Day 0 | X | X | X | X | X | X | X | x | X | X | x | X | X | X | X | X | X | X |
| | | Week 3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| xxxxxx | xxxxxxxxx | Day 0 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х | X | X | x |
| | | Week 3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ••• | | | | | | | | | | | | | | | | | | | | |

path\l\_program.sas date time

Programming note: Sort by subject ID.

Programming note: provide a key cover sheet for all the columns.

Allakos, Inc. AK001-002

Listing 16.2.6.21.8.3 36-Item Short Form Health Survey (SF-36) Part 3 of 3

| Subject ID | Treatment Group | Target Visit | VT4 | SF2 | GH2 | GH3 | GH4 | GH5 | Total Score |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXXXXX | Day 0 | X | X | X | X | X | X | XX |
| | | Week 3 | X | X | X | X | X | X | XX |
| | | ••• | | | | | | | |
| XXXXXX | XXXXXXXXX | Day 0 | X | X | X | X | X | X | XX |
| | | Week 3 | X | X | X | X | X | X | XX |
| xxxxxx | xxxxxxxxx | Day 0 | X | X | X | X | X | X | XX |
| | | Week 3 | X | X | X | X | X | X | XX |
| xxxxxx | xxxxxxxxx | Day 0 | X | X | X | X | X | X | XX |
| | | Week 3 | X | X | X | X | X | X | XX |

path\l\_program.sas date time

Programming note: Sort by subject ID.

Programming note: provide a key cover sheet for all the columns.

Programming note: Repeat listing for the listing listed below---

Listing 16.2.6.21.9 Asthma Control Test (ACT) {Replace item name columns with columns "ACT1", "ACT2", "ACT3",

"ACT4", and "ACT5"}

Listing 16.2.6.21.10 Spirometry Test

| | Treatment | | | Date Performed | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Group | Target Visit | Performed? | (Study Day) | Time | FEV1(%) | FVC(%) | FEF(%) |
| XXXXXX | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | XX | XX | XX |
| | | Week 3 | Yes/No | date9. (xx) | time5. | XX | XX | XX |
| | | Week 7 | Yes/No | date9. (xx) | time5. | XX | XX | XX |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | XX | XX | xx |
| | | Week 3 | Yes/No | date9. (xx) | time5. | XX | XX | XX |
| | | Week 7 | Yes/No | date9. (xx) | time5. | xx | XX | XX |

Note: Study day is calculated as days since the date of first dose of study drug. FEV1=Forced Expiratory Volume in 1 Second; FVC=Forced Vital Capacity; FEF=Forced Expiratory Flow

path\l program.sas date time

Listing 16.2.6.21.11.1 Sub-study Biomarkers Part 1 of 2

| | Treatment | Target | Collection Date | Collection | | | | | | Ca | arboxypeptida | se |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Group | Visit | (Study Day) | Time | ECP | Histamin | Tryptase | Prostaglandins | Leukotrienes | Chymase | A3 | Cytokines |
| | | ъ . | 1.0() | | | | | | | | | |
| XXXXXX | XXXXXXXXX | Day -3 | date9. (xx) | time5. | X | X | X | X | X | X | X | X |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | |
| xxxxxx | xxxxxxxxx | Day -3 | date9. (xx) | time5. | x | X | x | X | X | X | X | X |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X |
| xxxxxx | xxxxxxxxx | Day -3 | date9. (xx) | time5. | X | X | X | X | X | X | X | x |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | |
| xxxxxx | xxxxxxxxx | Day -3 | date9. (xx) | time5. | X | X | x | X | X | X | X | x |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | |
| ••• | | | | | | | | | | | | |

Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Listing 16.2.6.21.11.2 Sub-study Biomarkers Part 2 of 2

| Subject ID | Treatment<br>Group | Target<br>Visit | Collection Date<br>(Study Day) | Collection<br>Time | IL-5 | IL-17 | IFN | IL-4 | IL-13 | TSLP | IL-33 | IL-8 | TNF | Albumin | MPO | Growth<br>Factors |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx | Day -3 | date9. (xx) | time5. | X | X | x | x | x | X | x | x | X | X | x | X |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | | | | | |
| XXXXXX | xxxxxxxxx | Day -3 | date9. (xx) | time5. | X | X | x | X | x | x | x | X | X | X | X | X |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | | | | | |
| XXXXXX | xxxxxxxxx | Day -3 | date9. (xx) | time5. | X | X | x | X | X | X | X | X | X | X | X | X |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | ••• | | | | | | | | | | | | | | |
| xxxxxx | xxxxxxxxx | Day -3 | date9. (xx) | time5. | X | X | x | x | x | x | x | X | X | X | x | x |
| | | Week 2 | date9. (xx) | time5. | X | X | X | X | X | X | X | X | X | X | X | X |
| | | • • • | | | | | | | | | | | | | | |
| • • • | | | | | | | | | | | | | | | | |

Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Programming note: Sort by subject ID. Listing will include all the biomarkers from biomarker analysis.

Programming note: Please be sure all biomarkers are listed. The column headings need to be inserted based on the actual data to be received.

**Listing 16.2.7.22.1** Adverse Events

| | | | | Start | End | Start after last | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 5 | | | E Verbatim Term // | Date/Time <sup>[1]</sup> | Date/Time <sup>[1]</sup> | visit? | | | Relationship | Action Taken | Other | |
| ID | Group | # | Preferred Term | (Study Day) | (Study Day) | If Yes, Visit Date? | Serious | Severity | to Study Drug | with Study Drug | Action | Outcome |
| | | 1 | Manhatina Tama // | 1-4-0 /tim-5 | 1-4-0 /tim-5 | Yes/Date9. | Var/Na | | | | | |
| XXXXXX | xxxxxxxxx | 1 | Verbatim Term // Preferred Term | date9./time5. | date9./time5. | res/Date9. | Yes/No | severity | relationship | action | action | outcome |
| | | 2 | Verbatim Term // | (xx)<br>date9./time5. | (xx) date9./time5. | No/ | Yes/No | aarramitr. | relationship | action | action | outoom o |
| | | 2 | Preferred Term | | | 110/ | I CS/INO | severity | relationship | action | action | outcome |
| | | 2 | Verbatim Term // | (xx)<br>date9./time5. | (xx) date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome |
| | | 3 | Preferred Term | (xx) | (xx) | i es/Date9. | I CS/INO | severity | relationship | action | action | outcome |
| | | | riciciica i ciiii | (XX) | (XX) | | | | | | | |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | • | • | | | |
| | | 2 | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | | | | | |
| | | 3 | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | | | | | |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome |
| | MAMMAMA | • | Preferred Term | (xx) | (xx) | 1 co/ Date). | 1 05/110 | severity | relationship | action | uction | outcome |
| | | 2. | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | - 121 | | 20.0110 | | | | |
| | | 3 | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | | <b>.</b> | | | |
| XXXXXX | xxxxxxxxx | 1 | Verbatim Term // | date9./time/5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | | | | | |
| | | 2 | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | | | | | |
| | | 3 | Verbatim Term // | date9./time/5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome |
| | | | Preferred Term | (xx) | (xx) | | | | | | | |
| • • • | | | | | | | | | | | | |

\* Pre-treatment adverse event
# Post-treatment adverse event
[1] If time is marked unknown fill the time with "Unk", otherwise with "--"
Note: Study day is calculated as days since the date of first dose of study drug.

| path\l_program.sas date time<br>Programming note: sort by subject | ach subject. Please ensure ALL data from AE CRF appear in listing. |
|---|---|

Listing 16.2.7.22.2
Treatment-Emergent Serious Adverse Events (Collected on AE CRF)

| Subject | Treatment | AE | Verbatim Term // | Start Date | Start | End Date | End | | Relationship | Action Taken with Study | Other | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Group | # | Preferred Term | (Study Day) | Time | (Study Day) | Time | Severity | to Study Drug | Drug | Action | Outcome |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 2 | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 3 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 2 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 3 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 2 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 3 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| xxxxxx | xxxxxxxxx | 1 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 2 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |
| | | 3 | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome |

Note: Study day is calculated as days since the date of first dose of study drug. path\l program.sas date time

Programming note: sort by subject ID and onset date and resolution date within each subject.

Programming note: Repeat listing for the following:

Listing 16.2.7.22.3 Fatal Treatment-Emergent Serious Adverse Events (Collected on AE CRF)

Listing 16.2.7.22.4 Non-Fatal Treatment-Emergent Serious Adverse Events (Collected on AE CRF)

Listing 16.2.8.23.1.1 Central Laboratory Normal Ranges – Conventional Units

| | | Conventiona | al Units | System Internation | onal Units | |
|---|---|---|---|---|---|---|
| Panel Name | Laboratory Test | Normal Range | Unit | Normal Range | Unit | Effective Date |
| Hematology | WBC<br>Hematocrit<br>Hemoglobin | min-max<br>min-max<br>min-max | unit.<br>unit.<br>unit. | min-max<br>min-max<br>min-max | unit.<br>unit.<br>unit. | date9.<br>date9.<br>date9. |
| Serum Chemistry | AST | min-max | unit. | min-max | unit. | date9. |
| Urinalysis | <br>рН<br> | min-max | unit. | min-max | unit. | date9. |

path\l\_program.sas date time

Programming note: listing will include all the laboratory tests with normal ranges in central lab data. Repeat for Listing 16.2.8.23.1.2 using SI Units

Allakos, Inc.

AK001-002

Listing 16.2.8.23.2.1 Hematology – Conventional Units Part 1 of 2

| Subject<br>ID | Treatment<br>Group | Target<br>Visit | Performed? | Collection<br>Date<br>(Study Day) | | WBC<br>(10 <sup>9</sup> /L) | Neutrophils (%) | Neutrophils<br>(10 <sup>9</sup> /L) | Lymphocytes (%) | Lymphocytes (10 <sup>9</sup> /L) | Monocytes<br>(%) | Monocytes (10 <sup>9</sup> /L) | Eosinophils (%) | Eosinophils (10 <sup>9</sup> /L) | Basophils (%) | Basophils<br>(10 <sup>9</sup> /L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Conconino | Yes/No | date9. (xx) | tim of | **** | | | *** | | | | | | **** | *** |
| XXXXXX | xxxxxxxxx | Screening | | ` ′ | time5. | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | XXXXXXXXX | Screening | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XX.XX | XX,XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX |
| xxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | XX.XX | xx.xx | xx.xx | XX.XX | xx.xx | XX,XX | xx.xx | XX.XX | XX.XX | xx.xx | xx.xx |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XX.XX | XX,XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XX.XX | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| • • • • | | | | | | | | | | | | | | | | |

Note; L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Listing 16.2.8.23.2.2 Hematology – Conventional Units Part 2 of 2

| Subject<br>ID | Treatment<br>Group | Target<br>Visit | Collection<br>Date<br>(Study Day) | Collection<br>Time | Platelets (10 <sup>9</sup> /L) | RBC<br>(10 <sup>12</sup> /L) | Hemoglobin (mg/dL) | Hematocrit (%) | Reticulocytes (10 <sup>9</sup> /L) | Reticulocytes (%) | MCV<br>(fL) | Heinz Bodies (10 <sup>9</sup> /L) | MCH<br>(pg) | MCHC<br>(g/dL) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VVVVVV | xxxxxxxxx | Screening | date9. (xx) | time5. | xxx | VV VV | VV V | VVV | VV V | XX.X | vvv | VVV | VV V | VVV |
| ΑΛΛΛΛΛ | ********* | • | ` ' | | | XX.XX | XX.X | XX.X | XX.X | | XX.X | XXX | XX.X | XX.X |
| | | Day -3 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | Week 2 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| xxxxxx | xxxxxxxxx | Screening | date9. (xx) | time5. | xxx | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | Day -3 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | xx.x | XX.X | XX.X | xxx | XX.X | XX.X |
| | | Week 2 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | ••• | | | | | | | | | | | | |
| xxxxxx | xxxxxxxxx | Screening | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | Day -3 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | Week 2 | date9. (xx) | time5. | xxx | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | | 1.40() | · · · · · · · | | | | | | | | | | |
| XXXXXX | xxxxxxxxx | Screening | ` ' | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | Day -3 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | Week 2 | date9. (xx) | time5. | XXX | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X | XXX | XX.X | XX.X |
| | | ••• | | | | | | | | | | | | |
| ••• | | | | | | | | | | | | | | |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug.

path\l program.sas date time

Programming note: Sort by subject ID. Listing will include all the laboratory tests from central lab data in Hematology, and conventional units will be displayed. Repeat for Listing 16.2.8.23.2.3 using SI Units

AK001-002

Listing 16.2.8.23.3.1 **Serum Chemistry – Conventional Units** Part 1 of 2

| Subject<br>ID | Treatment<br>Group | Target Visit I | Performed? | Collection<br>Date (Study<br>Day) | Collection<br>Time | ALT<br>(SGPT)<br>(U/L) | AST<br>(SGOT)<br>(U/L) | Alkaline<br>Phosphatase<br>(U/L) | GGT<br>(U/L) | Albumin<br>(g/dL) | Total<br>Bilirubin<br>(mg/dL) | Direct<br>Bilirubin<br>(mg/dL) | BUN<br>(mg/dL) | Creatinine (mg/dL) | Creatine<br>Kinase<br>(U/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | G | <b>3</b> 7 / <b>N</b> 1 . | 1-(-0 ( ) | 455 | | | | | | | | | | |
| XXXXXX | xxxxxxxxx | _ | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | x.x |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| xxxxxx | xxxxxxxxx | <br>Screening | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| ΛΛΛΛΛΛ | λλλλλλλλλλ | U | Yes/No | ` / | | | | | | | | | | | |
| | | Day -3 | | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| xxxxxx | xxxxxxxxx | | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | Day -3 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | Week 2 | Yes/No | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XX | X.X | X.X |
| | | ••• | | | | | | | | | | | | | |
| ••• | | | | | | | | | | | | | | | |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Listing 16.2.8.23.3.2 Serum Chemistry – Conventional Units Part 2 of 2

| xxxxxxx | Screening Day -3 Week 2 Screening Day -3 Week 2 | date9. (xx)<br>date9. (xx)<br>date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5.<br>time5.<br>time5. | xxx<br>xxx<br>xxx<br>xxx | X.X<br>X.X<br>X.X | xxx<br>xxx<br>xxx | xx<br>xx<br>xx<br>xx | xxx<br>xxx<br>xxx<br>xxx | XX.X<br>XX.X<br>XX.X |
|---|---|---|---|---|---|---|---|---|---|
| | Day -3<br>Week 2<br><br>Screening<br>Day -3 | date9. (xx)<br>date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5. | xxx<br>xxx<br>xxx | x.x<br>x.x | xxx<br>xxx<br>xxx | xx<br>xx<br>xx | xxx<br>xxx<br>xxx | XX.X<br>XX.X |
| xxxxxx | Week 2<br><br>Screening<br>Day -3 | date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5. | xxx<br>xxx | x.x<br>x.x | xxx<br>xxx | xx<br>xx | xxx<br>xxx | XX.X |
| xxxxxx | Screening<br>Day -3 | date9. (xx)<br>date9. (xx) | time5. | xxx | X.X | XXX | xx | xxx | |
| xxxxxx | Screening<br>Day -3 | date9. (xx) | | | | | | | XX.X |
| | Day -3 | date9. (xx) | | | | | | | |
| | - | ` / | | | X.X | XXX | XX | XXX | XX.X |
| | TT COR Z | date9. (xx) | time5. | xxx | X.X | XXX | xx | XXX | XX.X |
| xxxxxx | Screening | date9. (xx) | time5. | XXX | X.X | xxx | XX | XXX | XX.X |
| | Day -3 | date9. (xx) | time5. | XXX | X.X | XXX | XX | XXX | XX.X |
| | Week 2 | date9. (xx) | time5. | XXX | X.X | xxx | XX | XXX | xx.x |
| xxxxxx | Screening | date9. (xx) | time5. | XXX | X.X | xxx | xx | XXX | XX.X |
| | | date9. (xx) | time5. | XXX | X.X | XXX | XX | XXX | XX.X |
| | Week 2 | date9. (xx) | time5. | XXX | X.X | XXX | XX | XXX | xx.x |
| | | Day -3 Week 2 Screening Day 1 Week 2 | Day -3 date9. (xx) Week 2 date9. (xx) xxxxxx Screening date9. (xx) Day 1 date9. (xx) Week 2 date9. (xx) | Day -3 date9. (xx) time5. Week 2 date9. (xx) time5. Screening date9. (xx) time5. Day 1 date9. (xx) time5. Week 2 date9. (xx) time5. Week 2 date9. (xx) time5. | Day -3 date9. (xx) time5. xxx Week 2 date9. (xx) time5. xxx Screening date9. (xx) time5. xxx Day 1 date9. (xx) time5. xxx Week 2 date9. (xx) time5. xxx Xxx Xx | Day -3 date9. (xx) time5. xxx x.x x.x Week 2 date9. (xx) time5. xxx x.x x | Day -3 date9. (xx) time5. xxx xx xxx xxx xxx xxx xxx xxx xxx xx | Day -3 date9. (xx) time5. xxx x.x xxx xx | Day -3 date9. (xx) time5. xxx x |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Programming note: Sort by subject ID. Listing will include all the laboratory tests from central lab data in Serum Chemistry, and conventional units will be displayed. Repeat for Listing 16.2.8.23.3.3 using SI Units

Listing 16.2.8.23.4 Urinalysis

| | | | | Collection | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | Target | | Date (Study | Collection | Specific | | | | | | |
| ID | Group | Visit | Performed? | Day) | Time | Gravity | Color | Protein | рН | Blood | Glucose | Ketones |
| XXXXXX | XXXXXXXXX | Screening | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| | | Day -3 | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| | | Week 2 | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| MAMA | MAMMAM | Day -3 | Yes/No | date9. (xx) | time5. | result | result | result | | | result | result |
| | | Week 2 | Yes/No | date9. (xx) | time5. | result | result | result | | | result | result |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| | | Day -3 | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| | | Week 2 | Yes/No | date9. (xx) | time5. | result | result | result | | | result | result |
| xxxxxx | xxxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | result | result | result | result | result | result | result |
| ААААА | АХАХАХХХ | Day -3 | Yes/No | date9. (xx) | time5. | result | result | result | | | result | result |
| | | Week 2 | Yes/No | date9. (xx) | time5. | result | result | result | | | result | result |
| | | | 1 05/110 | uate). (AA) | times. | resurt | resurt | icsuit | icsuit | resurt | resurt | icsuit |
| | | ••• | | | | | | | | | | |
| ••• | | | | | | | | | | | | |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

Programming note: Sort by subject ID. Listing will include all the laboratory tests from central lab data in Urinalysis.

Programming note: Please be sure all lab parameters are listed. The column headings need to be inserted based on the actual data to be received.

Listing 16.2.8.24.1 Vital Signs

| Subject Treatment<br>ID Group | Target<br>Visit | Performed? | Date of<br>Measurement<br>(Study Day) | Start Time<br>Supine Position | Time of<br>Measurement | Height (cm) | Weight (kg) | Temperature (°C) | Respiration<br>Rate<br>(breaths/min) | Systolic<br>Blood Pressure<br>(mmHg) | Diastolic<br>Blood Pressure<br>(mmHg) | Pulse Rate<br>(beats/min) | Any Findings<br>Abnormal? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx xxxxxxxx | Screening | Yes/No | date9. (xx) | time5. | time5. | XX.X. | xxx.x | xx.x | xx | xxx | xxx | xx | Yes: CS/NCS /<br>No |
| | Day -3 | | date9. (xx) | time5. | time5. | | xxx.x | XX.X | xx | XXX | xxx | xx | Yes: CS/NCS /<br>No |
| | Day 0 Pre-<br>dose | | date9. (xx) | time5. | time5. | | XXX.X | XX.X | xx | xxx | xxx | XX | Yes: CS/NCS /<br>No |
| xxxxx xxxxxxxx | Screening | | date9. (xx) | time5. | time5. | XX.X. | xxx.x | xx.x | xx | xxx | xxx | xx | Yes: CS/NCS /<br>No |
| | Day -3 | | date9. (xx) | time5. | time5. | | xxx.x | XX.X | xx | XXX | xxx | xx | Yes: CS/NCS /<br>No |
| | Day 0 Pre-<br>dose | | date9. (xx) | time5. | time5. | | XXX.X | XX.X | xx | xxx | XXX | xx | Yes: CS/NCS /<br>No |
| xxxxxx xxxxxxxxx | Screening | | date9. (xx) | time5. | time5. | XX.X. | xxx.x | xx.x | xx | xxx | xxx | xx | Yes: CS/NCS /<br>No |
| | Day 1 Pre-<br>Dose | | date9. (xx) | time5. | time5. | | xxx.x | XX.X | xx | xxx | xxx | xx | Yes: CS/NCS /<br>No |
| | Week 2 | | date9. (xx) | time5. | time5. | | xxx.x | xx.x | XX | xxx | xxx | xx | Yes: CS/NCS /<br>No |

Note: CS= Clinically Significant; NCS = Not Clinically Significant; \*=Potentially Clinically Significant. On Days 0, 21 and 49, vital signs will be measured pre-dose, every 15 minutes after the start of infusion, and immediately following the end of infusion. Study day is calculated as days since the date of first dose of study drug.

path\l program.sas date time

Listing 16.2.8.24.2 Vital Sign Results of Potential Clinical Significance

| C. Live ID | Total Control | Demonstruction ( mid) | Cuit aui a | Target | Collection Date | | D 14 |
|---|---|---|---|---|---|---|---|
| Subject ID | Treatment Group | Parameter (unit) | Criteria | Visit | (Study Day) | Collection Time | Results |
| xxxxxx | xxxxxxxxx | Temperature (°C) | criteria | Week x | date9. (xx) | time5. | result |
| | | Systolic Blood<br>Pressure (mmHg) | criteria | Week x | date9. (xx) | time5. | result |
| xxxxxx | xxxxxxxxx | Temperature (°C) | criteria | Week x | date9. (xx) | time5. | result |
| | | Systolic Blood<br>Pressure (mmHg) | criteria | Week x | date9. (xx) | time5. | result |
| xxxxxx | xxxxxxxxx | Temperature (°C) | criteria | Week x | date9. (xx) | time5. | result |
| | | Systolic Blood<br>Pressure (mmHg) | criteria | Week x | date9. (xx) | time5. | result |

Note: CS= Clinically Significant; NCS = Not Clinically Significant. Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time